CLINICAL TRIAL: NCT03548207
Title: A Phase 1b-2, Open-Label Study of JNJ-68284528, A Chimeric Antigen Receptor T-Cell (CAR-T) Therapy Directed Against BCMA in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of JNJ-68284528, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against B-Cell Maturation Antigen (BCMA) in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: CARTITUDE-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108480; 68284528MMY2001 (Other: Janssen Research & Development, LLC); 2018-000121-32 (EudraCT Number)
Expanded Access: NCT05346835 (Available)
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-68284528 (Experimental): After lymphodepletion JNJ-68284528 will be administered as a single infusion.
  Interventions: Biological: JNJ-68284528

INTERVENTIONS:
Biological: JNJ-68284528 — JNJ-68284528 consist of autologous T lymphocytes transduced with LCAR-B38M, a lentiviral vector to express a chimeric antigen receptor targeting the human B cell maturation antigen (anti-BCMA CAR).

SUMMARY:
The purpose of the study is to characterize safety of JNJ-68284528 and establish the recommended Phase 2 dose (RP2D) (Phase 1b) and to evaluate the efficacy of JNJ-68284528 (Phase 2).

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of JNJ-68284528. The study will include two phases. In Phase1b the study will enroll adults with multiple myeloma with interval assessments for potential dose escalation or de-escalation in subsequent participants. The dose selected at the completion of phase 1b will be used in Phase 2. Following consent, enrolled participants will undergo an apheresis procedure to collect cells for manufacture of investigational drug product (JNJ-68284528). Following manufacture of the drug product, participants will undergo lymphodepletion prior to infusion of JNJ-68284528. Participants will be followed for at least 2 years after study drug infusion, with long-term 15 year follow-up on a separate study. The study will evaluate safety, biomarkers, pharmacokinetic/pharmacodynamic evaluations and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Have documented diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Have measurable disease at Screening as defined by any of the following a) Serum monoclonal paraprotein (M-protein) level more than or equal to (>=) 1.0 gram per deciliter(g/dL) or urine M-protein level >=200 milligram per 24 hours (mg/24hr); or b) Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin free light chain 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Have received at least 3 prior multiple myeloma treatment lines of therapy or are double refractory to an immunomodulatory drug (IMiD) and proteasome inhibitor (PI) (refractory multiple myeloma as defined by IMWG consensus criteria). Note: induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single lines of therapy a) Undergone at least 1 complete cycle of treatment for each line of therapy, unless progressive disease (PD) was the best response to the regimen
* Have received as part of previous therapy a PI, an IMiD, and an anti-CD38 antibody
* Participant must have documented evidence of progressive disease based on investigator's determination of response by the IMWG criteria on or within 12 months of their last line of therapy. Confirmation may be from either central or local testing. Also, participants with documented evidence of progressive disease (as above) within the previous 6 months and who are refractory or non-responsive to their most recent line of therapy afterwards are eligible
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1

Exclusion Criteria:

* Have received prior treatment with chimeric antigen receptor T (CAR-T) therapy directed at any target
* Have received any therapy that is targeted to B-cell maturation antigen (BCMA)
* Have following cardiac conditions: a) New York Heart Association (NYHA) stage III or IV congestive heart failure b) Myocardial infarction or coronary artery bypass graft (CABG) less than or equal to (<=) 6 months prior to enrollment c) History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration d) History of severe non-ischemic cardiomyopathy e) Impaired cardiac function (left ventricular ejection fraction [LVEF] less than [<]45%) as assessed by echocardiogram or multiple-gated acquisition (MUGA) scan (performed less than or equal to (<=) 8 weeks of apheresis)
* Received a cumulative dose of corticosteroids equivalent to >= 70 mg of prednisone within the 7 days prior to apheresis
* Have received either of the following: a) An allogenic stem cell transplant within 6 months before apheresis. Participants who received an allogeneic transplant must be off all immunosuppressive medications for 6 weeks without signs of graft-versus-host disease (GVHD) b) An autologous stem cell transplant less than or equal to (<=) 12 weeks before apheresis
* Have known active, or prior history of central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- United States (17):
  - Mayo Clinic Cancer Center-Scottsdale, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Froedtert Memorial, Milwaukee, Wisconsin
- Japan (4):
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nagoya City University Hospital, Nagoya
  - Hokkaido University Hospital, Sapporo
  - Japanese Red Cross Medical Center, Shibuya City

REFERENCES:
- [Derived] Lopez-Munoz N, Bar N, Diels J, van Sanden S, Mendes J, Lee S, Hernando T, Lendvai N, Patel N, Ishida T, Er J, Harrison SJ. Ciltacabtagene Autoleucel Versus Idecabtagene Vicleucel in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma with 2-4 Prior Lines of Therapy: Updated Matching-Adjusted Indirect Comparison. Adv Ther. 2026 Feb 2. doi: 10.1007/s12325-025-03479-y. Online ahead of print. PMID 41627370
- [Derived] Jagannath S, Martin TG, Lin Y, Cohen AD, Raje N, Htut M, Deol A, Agha M, Berdeja JG, Lesokhin AM, Liegel JJ, Rossi A, Lieberman-Cribbin A, Usmani SZ, Dhakal B, Parekh S, Li H, Wang F, Montes de Oca R, Plaks V, Sun H, Banerjee A, Schecter JM, Lendvai N, Madduri D, Lengil T, Zhu J, Koneru M, Akram M, Patel N, Costa Filho O, Jakubowiak AJ, Voorhees PM. Long-Term (>/=5-Year) Remission and Survival After Treatment With Ciltacabtagene Autoleucel in CARTITUDE-1 Patients With Relapsed/Refractory Multiple Myeloma. J Clin Oncol. 2025 Sep;43(25):2766-2771. doi: 10.1200/JCO-25-00760. Epub 2025 Jun 3. PMID 40459151
- [Derived] Palmer S, Lin Y, Martin TG, Jagannath S, Jakubowiak A, Usmani SZ, Buyukkaramikli N, Phelps H, Slowik R, Pan F, Valluri S, Pacaud L, Jackson G. Extrapolation of Survival Data Using a Bayesian Approach: A Case Study Leveraging External Data from Cilta-Cel Therapy in Multiple Myeloma. Oncol Ther. 2023 Sep;11(3):313-326. doi: 10.1007/s40487-023-00230-x. Epub 2023 Jun 4. PMID 37270762
- [Derived] Raghunandan S, Pauly M, Blum WG, Qayed M, Dhodapkar MV, Elkhalifa M, Watkins B, Schoettler M, Horwitz E, Parikh S, Chandrakasan S, Leung K, Bryson E, Deeb L, Kaufman JL, Worthington-White D, Alazraki A, Schecter JM, Madduri D, Jackson CC, Zudaire E, Taraseviciute-Morris A, Babich A, Nesheiwat T, Vogel M, Lendvai N, Pacaud L, Williams KM. BCMA CAR-T induces complete and durable remission in refractory plasmablastic lymphoma. J Immunother Cancer. 2023 May;11(5):e006684. doi: 10.1136/jitc-2023-006684. PMID 37137553
- [Derived] Mateos MV, Weisel K, Martin T, Berdeja JG, Jakubowiak A, Stewart AK, Jagannath S, Lin Y, Diels J, Ghilotti F, Thilakarathne P, Perualila NJ, Cabrieto J, Haefliger B, Erler-Yates N, Hague C, Jackson CC, Schecter JM, Strulev V, Nesheiwat T, Pacaud L, Einsele H, Moreau P. Adjusted comparison of outcomes between patients from CARTITUDE-1 versus multiple myeloma patients with prior exposure to proteasome inhibitors, immunomodulatory drugs and anti-CD38 antibody from the prospective, multinational LocoMMotion study of real-world clinical practice. Haematologica. 2023 Aug 1;108(8):2192-2204. doi: 10.3324/haematol.2022.280482. PMID 36546453
- [Derived] Cohen AD, Hari P, Htut M, Berdeja JG, Usmani SZ, Madduri D, Olyslager Y, Goldberg JD, Schecter JM, Jackson CC, Gries KS, Fastenau JM, Valluri S, Deraedt W, Akram M, Crawford R, Morrison R, Doward L, Morgan K, Seldam ST, Jakubowiak A, Jagannath S. Patient Perceptions Regarding Ciltacabtagene Autoleucel Treatment: Qualitative Evidence From Interviews With Patients With Relapsed/Refractory Multiple Myeloma in the CARTITUDE-1 Study. Clin Lymphoma Myeloma Leuk. 2023 Jan;23(1):68-77. doi: 10.1016/j.clml.2022.10.001. Epub 2022 Oct 11. PMID 36357295
- [Derived] Martin T, Lin Y, Agha M, Cohen AD, Htut M, Stewart AK, Hari P, Berdeja JG, Usmani SZ, Yeh TM, Olyslager Y, Goldberg JD, Schecter JM, Madduri D, Jackson CC, Deraedt W, Gries KS, Fastenau JM, Trudeau JJ, Akram M, Pacaud L, Jakubowiak A, Jagannath S. Health-related quality of life in patients given ciltacabtagene autoleucel for relapsed or refractory multiple myeloma (CARTITUDE-1): a phase 1b-2, open-label study. Lancet Haematol. 2022 Dec;9(12):e897-e905. doi: 10.1016/S2352-3026(22)00284-8. Epub 2022 Oct 7. PMID 36215989
- [Derived] Wu LS, Su Y, Li C, Zhou W, Jackson CC, Sun YN, Zhou H. Population-based cellular kinetic characterization of ciltacabtagene autoleucel in subjects with relapsed or refractory multiple myeloma. Clin Transl Sci. 2022 Dec;15(12):3000-3011. doi: 10.1111/cts.13421. Epub 2022 Oct 6. PMID 36204820
- [Derived] Martin T, Usmani SZ, Berdeja JG, Agha M, Cohen AD, Hari P, Avigan D, Deol A, Htut M, Lesokhin A, Munshi NC, O'Donnell E, Stewart AK, Schecter JM, Goldberg JD, Jackson CC, Yeh TM, Banerjee A, Allred A, Zudaire E, Deraedt W, Olyslager Y, Zhou C, Pacaud L, Madduri D, Jakubowiak A, Lin Y, Jagannath S. Ciltacabtagene Autoleucel, an Anti-B-cell Maturation Antigen Chimeric Antigen Receptor T-Cell Therapy, for Relapsed/Refractory Multiple Myeloma: CARTITUDE-1 2-Year Follow-Up. J Clin Oncol. 2023 Feb 20;41(6):1265-1274. doi: 10.1200/JCO.22.00842. Epub 2022 Jun 4. PMID 35658469
- [Derived] Van Oekelen O, Aleman A, Upadhyaya B, Schnakenberg S, Madduri D, Gavane S, Teruya-Feldstein J, Crary JF, Fowkes ME, Stacy CB, Kim-Schulze S, Rahman A, Lagana A, Brody JD, Merad M, Jagannath S, Parekh S. Neurocognitive and hypokinetic movement disorder with features of parkinsonism after BCMA-targeting CAR-T cell therapy. Nat Med. 2021 Dec;27(12):2099-2103. doi: 10.1038/s41591-021-01564-7. Epub 2021 Dec 10. PMID 34893771
- [Derived] Berdeja JG, Madduri D, Usmani SZ, Jakubowiak A, Agha M, Cohen AD, Stewart AK, Hari P, Htut M, Lesokhin A, Deol A, Munshi NC, O'Donnell E, Avigan D, Singh I, Zudaire E, Yeh TM, Allred AJ, Olyslager Y, Banerjee A, Jackson CC, Goldberg JD, Schecter JM, Deraedt W, Zhuang SH, Infante J, Geng D, Wu X, Carrasco-Alfonso MJ, Akram M, Hossain F, Rizvi S, Fan F, Lin Y, Martin T, Jagannath S. Ciltacabtagene autoleucel, a B-cell maturation antigen-directed chimeric antigen receptor T-cell therapy in patients with relapsed or refractory multiple myeloma (CARTITUDE-1): a phase 1b/2 open-label study. Lancet. 2021 Jul 24;398(10297):314-324. doi: 10.1016/S0140-6736(21)00933-8. Epub 2021 Jun 24. PMID 34175021

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As planned, data for Phase 2 participants were reported separately for US population (78 participants) and Japan population (13 participants).
Groups:
- Phase 1b (US Population): Participants received a conditioning regimen of cyclophosphamide 300 milligrams per meter square (mg/m^2) intravenous (IV) infusion and fludarabine 30 mg/m^2 as IV infusion daily for 3 days from Day -5 to Day -3. On Day 1, participants received target dose of JNJ-68284528 0.75*10^6 chimeric antigen receptor T (CAR-T) cells per kilogram (cells/kg) (range: 0.5-1.0*10^6 CAR-positive viable cells/kg) as IV infusion.
- Phase 2 (US Population): Participants received a conditioning regimen of cyclophosphamide 300 mg/m^2 IV infusion and fludarabine 30 mg/m^2 IV infusion daily for 3 days from Day -5 to Day -3. On Day 1, participants received recommended phase 2 dose (RP2D) dose of JNJ-68284528 0.75*10^6 CAR positive viable T cells/kg as IV infusion.
- Phase 2 (Japan Population): Participants received a conditioning regimen of cyclophosphamide 300 mg/m^2 IV infusion and fludarabine 30 mg/m^2 IV infusion daily for 3 days from Day -5 to Day -3. On Day 1, participants received RP2D dose of JNJ-68284528 0.75*10^6 CAR positive viable T cells/kg as IV infusion.
Period: Overall Study
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Started | 35 | 78 | 13
Treated | 29 | 68 | 9
Completed | 0 | 0 | 0
Not Completed | 35 | 78 | 13
Not completed — Death | 10 | 23 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Sponsor decision | 19 | 40 | 6
Not completed — Randomized but not treated | 6 | 10 | 4

BASELINE CHARACTERISTICS:
Population: All treated analysis set included all participants who received JNJ-68284528 infusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population) | Total
Number analyzed (Participants) | 29 | 68 | 9 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (6.42) | 62.5 (9.09) | 58.9 (8.87) | 61.7 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 25 | 4 | 44
  Male | 14 | 43 | 5 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 9 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 5 | 12 | 0 | 17
  White | 20 | 49 | 0 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 0 | 0 | 9 | 9
  United States | 29 | 68 | 0 | 97

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Adverse Events as Per Severity
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Time Frame: Day 1 up to 45.2 months
Population: All treated analysis set included all participants who received JNJ-68284528 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b (US Population)
Number analyzed (Participants) | 29
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 2
  Grade 4 | 26
  Grade 5 | 1

2. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved partial response (PR) or better according to international myeloma working group (IMWG) criteria. IMWG criteria for PR: greater than or equal to (>=) 50 percent (%) reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to less than (<) 200 milligrams (mg) per 24 hours. If the serum and urine M-protein were not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels was required in place of the M-protein criteria. If serum and urine M-protein were not measurable, and serum free light assay was also not measurable, >=50% reduction in bone marrow plasma cells (PCs) was required in place of M-protein, provided baseline bone marrow PC percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: Day 1 up to 45.2 months
Population: Modified intent-to-treat (mITT) analysis set included all participants who received a JNJ-68284528 infusion at the targeted recommended phase 2 dose (RP2D) dose level. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 68 | 8
Percentage of participants | 97.1 [89.8 to 99.6] | 100.0 [66.4 to 100.0]

3. Secondary Outcome: Phase 2: Number of Participants With Adverse Events (AEs) as Per Severity
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Severity was graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Time Frame: Day 1 up to 45.2 months
Population: All treated analysis set included all participants who received JNJ-68284528 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 68 | 9
Participants
  Grade 1 | 0 | 0
  Grade 2 | 0 | 1
  Grade 3 | 5 | 0
  Grade 4 | 58 | 8
  Grade 5 | 5 | 0

4. Secondary Outcome: Phase 1b and Phase 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-68284528 Transgene
Description: Maximum observed plasma concentration (Cmax) of JNJ-68284528 transgene was reported. Cmax was calculated in copies per microgram (mcg) genomic deoxyribonucleic acid (DNA).
Time Frame: Pre and post dose on Day 1, and Days 2, 3, 7, 10, 14, 21, 28, 42, 56, 78, 100, then every 4 weeks up to 1 year, and at the time of progressive disease or at study completion for participants without progressive disease (up to approximately 2.5 years)
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Mean (Standard Deviation); unit: copies per mcg genomic DNA
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
copies per mcg genomic DNA | 38965 (19408) | 52841 (29021) | 44077 (39911)

5. Secondary Outcome: Phase 1b and Phase 2: Actual Sampling Time of Last Measurable Analyte Concentration (Tlast) of JNJ-68284528 Transgene
Description: Tlast was defined as actual sampling time of last measurable (non-below quantification limit [BQL]) analyte concentration of JNJ-68284528 transgene.
Time Frame: Pre and post dose on Day 1 and Days 2, 3, 7, 10, 14, 21, 28, 42, 56, 78, 100, then every 4 weeks up to 1 year, and at the time of progressive disease or at study completion for participants without progressive disease (up to approximately 2.5 years)
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Days | 127.13 [26.15 to 715.00] | 122.98 [20.04 to 910.92] | 129.89 [24.97 to 568.92]

6. Secondary Outcome: Phase 1b and Phase 2: Area Under the Plasma Concentration Versus Time Curve From Time 0 To Last Measurable Concentration (AUC0-last) of JNJ-68284528 Transgene
Description: Area under the plasma concentration versus time curve from time 0 to last measurable concentration of JNJ-68284528 transgene was reported.
Time Frame: Pre and post dose on Day 1; Days 2, 3, 7, 10, 14, 21, 28, 42, 56, 78, 100, then every 4 weeks up to 1 year, and at the time of progressive disease or at study completion for participants without progressive disease (up to approximately 2.5 years)
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Mean (Standard Deviation); unit: Day*copies per mcg genomic DNA
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Day*copies per mcg genomic DNA | 588162 (466441) | 1356191 (1673474) | 4062950 (7293651)

7. Secondary Outcome: Phase 1b and Phase 2: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinite Time (AUC0-infinity) of JNJ-68284528 Transgene
Description: Area under the plasma concentration versus time curve from time 0 to infinite time of JNJ-68284528 transgene was reported.
Time Frame: as for outcome 5
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Day*copies per mcg genomic DNA
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 11 | 33 | 3
Day*copies per mcg genomic DNA | 542728 (345847) | 1321427 (1513726) | 7173538 (12191640)

8. Secondary Outcome: Phase 1b and Phase 2: Maximum Observed Plasma Concentration (Cmax) of CD3+CAR+ Cells in Blood After a Single Infusion of JNJ-68284528
Description: Maximum observed plasma concentration (Cmax) of CD3+CAR+ Cells was reported. Cmax was calculated in cells per microliter.
Time Frame: as for outcome 5
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Cells per microliter | 483 (464) | 1472 (2085) | 1614 (3718)

9. Secondary Outcome: Phase 1b and Phase 2: T Cell Persistence After a Single Infusion of JNJ-68284528
Description: T Cell persistence after a single infusion of JNJ-68284528 was reported. T Cell persistence was defined as actual sampling time of last measurable (non-below quantification limit [BQL]) analyte concentration.
Time Frame: as for outcome 5
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Days | 84.08 [12.89 to 715.00] | 100.23 [20.04 to 910.92] | 56.81 [12.72 to 568.92]

10. Secondary Outcome: Phase 1b and Phase 2: Area Under the Plasma Concentration Versus Time Curve From Time 0 To Last Measurable Concentration (AUC0-last) of CD3+CAR+ Cells in Blood After a Single Infusion of JNJ-68284528
Description: Area under the plasma concentration versus time curve from time 0 to last measurable concentration of CD3+CAR+ Cells was reported.
Time Frame: as for outcome 5
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Mean (Standard Deviation); unit: Day*cells per microliter
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Day*cells per microliter | 7758 (7599) | 40073 (79603) | 152904 (361949)

11. Secondary Outcome: Phase 1b and Phase 2: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinite Time (AUC0-infinity) of CD3+CAR+ Cells in Blood After a Single Infusion of JNJ-68284528
Description: Area under the plasma concentration versus time curve from time 0 to infinite time of CD3+CAR+ Cells in blood after a single infusion of JNJ-68284528 was reported.
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days*cells per microliter
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 11 | 33 | 2
Days*cells per microliter | 10937 (8658) | 31966 (58976) | 7144.5 (5905)

12. Secondary Outcome: Phase 1b and Phase 2: Mean Concentration of Soluble B-cell Maturation Antigen (BCMA) Levels in Serum After Single Infusion of JNJ-68284528
Description: Mean concentration of soluble BCMA levels in serum after single infusion of JNJ-68284528 were reported.
Time Frame: Days 352 and 1024
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure. Zero (0) participants in the number analyzed field for arm "Phase 2 (Japan Population)" at Day 1024 signifies that no participants were available for the analysis because no sBCMA samples were collected and analyzed due to change in planned analysis.
Measure: Mean (Full Range); unit: Micrograms per liter (mcg/L)
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 11 | 33 | 8
Micrograms per liter (mcg/L)
  Day 352 | 2.25 [NA to 7.65] — Here, "NA" signifies that lower limit of full range could not be estimated as it was below the quantification limit. | 2.01 [NA to 10.40] — Here, "NA" signifies that lower limit of full range could not be estimated as it was below the quantification limit. | 5.61 [NA to 23.0] — Here, "NA" signifies that lower limit of full range could not be estimated as it was below the quantification limit.
  Day 1024: number analyzed (Participants) | 11 | 33 | 0
  Day 1024 | 6.70 [0.31 to 14.7] | 7.05 [3.21 to 11.90] |

13. Secondary Outcome: Number of Participants With Depletion of BCMA Expressing Cells
Description: Number of participants with depletion of BCMA expressing cells were reported.
Time Frame: Pre dose (Day 1) up to 2 years
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure. Due to change in planned analysis, data was not collected and analyzed for "Phase 2 (Japan Population)" in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 0
Participants | 0 | 0 |

14. Secondary Outcome: Phase 1b and Phase 2: Serum Systemic Cytokine Concentrations
Description: Serum systemic cytokine concentrations (Interleukin [IL]-6, IL-10, and Interferon Gamma [IFN-g]) were reported.
Time Frame: Pre-infusion and 2 hours post infusion on Day 1, Days 2, 3, 7, 10, 14, 21, 28, 42, 56, 78, 100
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here 'n' (number analyzed) signifies participants who were evaluable at specified time points for specified categories.
Measure: Mean (Standard Error); unit: nanograms per liter
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
nanograms per liter
  Interleukin 6: Day 1 (Pre-infusion): number analyzed (Participants) | 29 | 67 | 9
  Interleukin 6: Day 1 (Pre-infusion) | 3.66 (4.280) | 3.81 (4.231) | 1.62 (1.597)
  Interleukin 6: Day 1 (2 hours post-infusion): number analyzed (Participants) | 23 | 31 | 9
  Interleukin 6: Day 1 (2 hours post-infusion) | 3.59 (3.892) | 4.05 (4.158) | 1.76 (1.602)
  Interleukin 6: Day 2: number analyzed (Participants) | 1 | 65 | 9
  Interleukin 6: Day 2 | 4.62 | 6.47 (6.783) | 2.74 (2.268)
  Interleukin 6: Day 3: number analyzed (Participants) | 29 | 67 | 9
  Interleukin 6: Day 3 | 7.31 (12.849) | 25.57 (110.008) | 3.87 (4.360)
  Interleukin 6: Day 7: number analyzed (Participants) | 27 | 65 | 9
  Interleukin 6: Day 7 | 25.43 (68.141) | 200.93 (434.850) | 128.50 (367.531)
  Interleukin 6: Day 10: number analyzed (Participants) | 29 | 67 | 9
  Interleukin 6: Day 10 | 247.99 (464.936) | 227.01 (405.250) | 108.05 (171.088)
  Interleukin 6: Day 14: number analyzed (Participants) | 28 | 67 | 9
  Interleukin 6: Day 14 | 42.03 (63.840) | 110.94 (512.499) | 20.62 (17.898)
  Interleukin 6: Day 21: number analyzed (Participants) | 27 | 68 | 9
  Interleukin 6: Day 21 | 227.45 (989.332) | 69.33 (291.552) | 14.25 (15.439)
  Interleukin 6: Day 28: number analyzed (Participants) | 27 | 64 | 9
  Interleukin 6: Day 28 | 67.89 (129.381) | 110.86 (593.155) | 18.73 (26.593)
  Interleukin 6: Day 42: number analyzed (Participants) | 28 | 61 | 9
  Interleukin 6: Day 42 | 56.16 (153.528) | 141.33 (908.434) | 12.23 (10.830)
  Interleukin 6: Day 56: number analyzed (Participants) | 27 | 64 | 9
  Interleukin 6: Day 56 | 12.44 (34.311) | 113.28 (749.566) | 8.12 (8.594)
  Interleukin 6: Day 78: number analyzed (Participants) | 29 | 62 | 9
  Interleukin 6: Day 78 | 56.25 (164.152) | 137.01 (753.322) | 3.91 (6.280)
  Interleukin 6: Day 100: number analyzed (Participants) | 24 | 65 | 9
  Interleukin 6: Day 100 | 2.36 (1.680) | 239.64 (1491.202) | 1.45 (1.123)
  Interleukin 10: Day 1 (pre-infusion): number analyzed (Participants) | 29 | 67 | 9
  Interleukin 10: Day 1 (pre-infusion) | 1.19 (1.170) | 1.68 (2.749) | 1.07 (0.795)
  Interleukin 10: Day 1 (2 hours post-infusion): number analyzed (Participants) | 26 | 31 | 9
  Interleukin 10: Day 1 (2 hours post-infusion) | 1.11 (0.924) | 1.94 (3.406) | 1.07 (0.795)
  Interleukin 10: Day 2: number analyzed (Participants) | 1 | 65 | 9
  Interleukin 10: Day 2 | 2.85 | 3.86 (6.114) | 1.90 (1.695)
  Interleukin 10: Day 3: number analyzed (Participants) | 29 | 67 | 9
  Interleukin 10: Day 3 | 2.65 (2.931) | 4.54 (8.318) | 2.10 (1.820)
  Interleukin 10: Day 7: number analyzed (Participants) | 27 | 65 | 9
  Interleukin 10: Day 7 | 27.95 (30.506) | 56.32 (81.383) | 89.21 (163.729)
  Interleukin 10: Day 10: number analyzed (Participants) | 29 | 67 | 9
  Interleukin 10: Day 10 | 36.44 (56.307) | 53.78 (156.803) | 102.71 (184.878)
  Interleukin 10: Day 14: number analyzed (Participants) | 28 | 66 | 9
  Interleukin 10: Day 14 | 20.50 (90.471) | 6.99 (15.549) | 6.20 (6.257)
  Interleukin 10: Day 21: number analyzed (Participants) | 27 | 68 | 9
  Interleukin 10: Day 21 | 5.14 (5.496) | 5.36 (14.437) | 1.06 (0.560)
  Interleukin 10: Day 28: number analyzed (Participants) | 27 | 64 | 9
  Interleukin 10: Day 28 | 2.30 (1.345) | 3.45 (6.740) | 2.19 (1.917)
  Interleukin 10: Day 42: number analyzed (Participants) | 28 | 61 | 9
  Interleukin 10: Day 42 | 2.36 (3.270) | 1.94 (2.682) | 1.52 (0.853)
  Interleukin 10: Day 56: number analyzed (Participants) | 27 | 64 | 9
  Interleukin 10: Day 56 | 2.17 (2.540) | 1.54 (0.967) | 2.38 (2.715)
  Interleukin 10: Day 78: number analyzed (Participants) | 29 | 62 | 9
  Interleukin 10: Day 78 | 1.84 (2.181) | 1.64 (1.499) | 1.08 (0.552)
  Interleukin 10: Day 100: number analyzed (Participants) | 24 | 65 | 9
  Interleukin 10: Day 100 | 1.45 (0.881) | 1.91 (1.920) | 0.72 (0.272)
  Interferon Gamma: Day1 (pre-infusion): number analyzed (Participants) | 29 | 67 | 9
  Interferon Gamma: Day1 (pre-infusion) | 13.37 (14.658) | 1.68 (2.749) | 25.29 (15.168)
  Interferon Gamma: Day1 (2 hours post-infusion): number analyzed (Participants) | 26 | 31 | 9
  Interferon Gamma: Day1 (2 hours post-infusion) | 21.68 (30.670) | 35.50 (53.105) | 25.29 (15.168)
  Interferon Gamma: Day 2: number analyzed (Participants) | 1 | 65 | 9
  Interferon Gamma: Day 2 | 50.87 | 3.86 (6.114) | 48.01 (30.732)
  Interferon Gamma: Day 3: number analyzed (Participants) | 29 | 67 | 9
  Interferon Gamma: Day 3 | 57.95 (59.699) | 4.54 (8.318) | 44.83 (48.154)
  Interferon Gamma: Day 7: number analyzed (Participants) | 27 | 65 | 9
  Interferon Gamma: Day 7 | 284.86 (397.735) | 56.32 (81.383) | 9043.92 (26714.417)
  Interferon Gamma: Day 10: number analyzed (Participants) | 29 | 67 | 9
  Interferon Gamma: Day 10 | 4095.68 (12586.211) | 53.78 (156.803) | 5351.97 (11598.493)
  Interferon Gamma: Day 14: number analyzed (Participants) | 28 | 66 | 9
  Interferon Gamma: Day 14 | 44.58 (41.813) | 6.99 (15.549) | 59.50 (48.748)
  Interferon Gamma: Day 21: number analyzed (Participants) | 27 | 68 | 9
  Interferon Gamma: Day 21 | 108.39 (113.492) | 5.36 (14.437) | 28.70 (22.852)
  Interferon Gamma: Day 28: number analyzed (Participants) | 27 | 64 | 9
  Interferon Gamma: Day 28 | 57.44 (82.982) | 3.45 (6.740) | 44.36 (45.668)
  Interferon Gamma: Day 42: number analyzed (Participants) | 28 | 61 | 9
  Interferon Gamma: Day 42 | 32.69 (39.456) | 1.94 (2.682) | 22.76 (22.233)
  Interferon Gamma: Day 56: number analyzed (Participants) | 27 | 64 | 9
  Interferon Gamma: Day 56 | 50.58 (143.096) | 1.54 (0.967) | 19.88 (32.794)
  Interferon Gamma: Day 78: number analyzed (Participants) | 29 | 62 | 9
  Interferon Gamma: Day 78 | 26.19 (34.120) | 1.64 (1.499) | 7.71 (4.433)
  Interferon Gamma: Day 100: number analyzed (Participants) | 24 | 65 | 9
  Interferon Gamma: Day 100 | 18.51 (18.052) | 1.91 (1.920) | 9.04 (4.958)

15. Secondary Outcome: Phase 1b and Phase 2: Maximum Observed Plasma Concentration (Cmax) of CAR-T Cells (CD3+CAR+ Cells in Blood) After a Single Infusion of JNJ-68284528
Description: Cmax of CAR-T cells (CD3+CAR+ cells in blood) after a single infusion of JNJ-68284528 was reported.
Time Frame: as for outcome 5
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Cells per microliter | 483 (464) | 1472 (2085) | 1614 (3718)

16. Secondary Outcome: Phase 1b and Phase 2: Maximum T Cell Expansion After a Single Infusion of JNJ-68284528
Description: Maximum T cell expansion was defined as maximum observed plasma concentration (Cmax) after a single Infusion of JNJ-68284528.
Time Frame: as for outcome 5
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Cells per microliter | 483 (464) | 1472 (2085) | 1614 (3718)

17. Secondary Outcome: Phase 1b and Phase 2: Percentage of Participants With Positive Antibodies to JNJ-68284528
Description: Percentage of participants with positive antibodies to JNJ-68284528 were reported.
Time Frame: Pre dose (Day 1) up to 2 years
Population: All treated analysis set included all participants who received JNJ-68284528 infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Percentage of participants | 48.3 | 35.3 | 44.4

18. Secondary Outcome: Phase 1b and Phase 2: Very Good Partial Response (VGPR) or Better Response Rate
Description: VGPR or better response rate was defined as the percentage of participants who achieved VGPR or complete response (CR) (including stringent complete response [sCR]) according to the IMWG criteria during or after the study treatment. VGPR: Serum and urine component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein level less than (<) 100 mg/24 hour; CR: negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% PCs in bone marrow; sCR: CR in addition to having a normal free light chain (FLC) ratio and an absence of clonal cells in bone marrow by immunohistochemistry, immunofluorescence, 2-4 color flow cytometry.
Time Frame: Pre dose (Day 1) up to 45.2 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 8
Percentage of participants | 96.6 [82.2 to 99.9] | 94.1 [85.6 to 98.4] | 100.0 [63.1 to 100.0]

19. Secondary Outcome: Phase 1b and Phase 2: Minimal Residual Disease (MRD) Negative Rate
Description: MRD negativity rate was defined as percentage of participants who had negative MRD by bone marrow aspirate at any timepoint after initial dose of JNJ-68284528 and before disease progression or starting subsequent therapy or retreatment with JNJ-68284528. MRD negativity rate was assessed by next-generation sequencing at a threshold of <10^5.
Time Frame: Pre dose (Day 1) up to 45.2 months
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here, N (number of participants analyzed) signifies participants with evaluable samples for MRD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 18 | 39 | 8
Percentage of participants | 100.0 [81.5 to 100.0] | 89.7 [75.8 to 97.1] | 75.0 [34.9 to 96.8]

20. Secondary Outcome: Phase 1b and Phase 2: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate was defined as the percentage of participants with best response of minimal response (MR) or better (including sCR, CR, VGPR, PR, and MR). MR was defined as >=25% but less than or equal to (<=) 49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50% to 89%. In addition to the above criteria, if present at baseline, >=50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: Pre dose (Day 1) up to 45.2 months
Population: mITT analysis Set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 9
Percentage of participants | 100.0 [88.1 to 100.0] | 97.1 [89.8 to 99.6] | 100.0 [63.1 to 100.0]

21. Secondary Outcome: Phase 1b and Phase 2: Duration of Response (DOR)
Description: DOR was defined as the time (in months) from the date of initial documented response (PR or better response) to the date of first documented evidence of progressive disease (PD) or death. PD is defined as an increase of 25% from the lowest response value in one of the following: serum and urine M-component (absolute increase must be >=0.5 gram per deciliter [g/dL] and >=200 mg/24 hours respectively); only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder, appearance of a new lesion(s), >=50% increase in circulating plasma cells if this was the only measure of disease.
Time Frame: Pre dose (Day 1) up to first documented PD or death (up to 45.2 months)
Population: Analysis population included responders (who achieved PR or better response) in mITT analysis set. mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 66 | 8
Months | NA [15.9 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [23.1 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [10.3 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

22. Secondary Outcome: Phase 1b and Phase 2: Time to First Response
Description: Time to first response was defined as the time between date of the initial infusion of JNJ-68284528 and the first efficacy evaluation that the participant met all criteria for PR or better. IMWG criteria for PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or <200 mg per 24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow PCs is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Pre dose (Day 1) up to 45.2 months
Population: Analysis population included responders in mITT analysis set. mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 66 | 8
Months | 0.95 [0.9 to 2.8] | 0.95 [0.9 to 10.7] | 0.92 [0.9 to 1.8]

23. Secondary Outcome: Phase 1b and Phase 2: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from the date of the initial infusion of JNJ-68284528 to the date of first documented disease progression.
Time Frame: Pre dose (Day 1) up to 45.2 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 8
Months | NA [16.79 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [24.08 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [11.17 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

24. Secondary Outcome: Phase 1b and Phase 2: Overall Survival
Description: Overall survival was defined as the time from the date of the initial infusion of JNJ-68284528 to the date of the participant's death.
Time Frame: Pre dose (Day 1) up to 45.2 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 29 | 68 | 8
Months | NA [27.24 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [32.20 to NA] — Here, NA signifies that median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 27.04 [18.40 to NA] — Here, NA signifies that upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

25. Secondary Outcome: Phase 2 (US Population): Change From Baseline in EuroQol Five Dimension Questionnaire (EQ-5D-5L) Utility Score at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Description: EQ-5D-5L was a 5-item questionnaire consisted of 2 components: a health state profile/a single utility index value and an optional VAS. EQ-5D health state profile/a single utility index value had 5 dimensions including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 response levels: 1 =no problems, 2 =slight problems, 3 =moderate problems, 4 =severe problems and 5 =extreme problems. The scores for the 5 dimensions were used to compute a single utility score ranging from 0 to 1 representing the general health status of the individual. Higher score indicated better health status. EQ-5D VAS was used to record participant's rating for his/her "health today" and ranging from 0 to 100, where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Population: mITT analysis Set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 54
Score on a scale
  Change at Day 7 | -0.1 [-0.1 to 0]
  Change at Day 28: number analyzed (Participants) | 53
  Change at Day 28 | 0 [-0.1 to 0]
  Change at Day 56: number analyzed (Participants) | 52
  Change at Day 56 | 0 [-0.1 to 0.1]
  Change at Day 78: number analyzed (Participants) | 46
  Change at Day 78 | 0 [0 to 0.1]
  Change at Day 100: number analyzed (Participants) | 49
  Change at Day 100 | 0 [0 to 0.1]
  Change at Day 128: number analyzed (Participants) | 40
  Change at Day 128 | 0 [0 to 0.1]
  Change at Day 156: number analyzed (Participants) | 36
  Change at Day 156 | 0 [0 to 0.1]
  Change at Day 184: number analyzed (Participants) | 40
  Change at Day 184 | 0 [0 to 0.1]
  Change at Day 212: number analyzed (Participants) | 33
  Change at Day 212 | 0.1 [0 to 0.1]
  Change at Day 240: number analyzed (Participants) | 32
  Change at Day 240 | 0.1 [0 to 0.1]
  Change at Day 268: number analyzed (Participants) | 36
  Change at Day 268 | 0.1 [0 to 0.1]
  Change at Day 296: number analyzed (Participants) | 33
  Change at Day 296 | 0.1 [0 to 0.1]
  Change at Day 324: number analyzed (Participants) | 14
  Change at Day 324 | 0 [0 to 0.1]
  Change at Day 352: number analyzed (Participants) | 7
  Change at Day 352 | 0.1 [0 to 0.2]
  Change at Day 380: number analyzed (Participants) | 2
  Change at Day 380 | -0.1 [-0.3 to 0.2]

26. Secondary Outcome: Phase 2 (Japan Population): Change From Baseline in EuroQol Five Dimension Questionnaire (EQ-5D-5L) Utility Score at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Description: as for outcome 25
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 8
Score on a scale
  Change at Day 7 | -0.05 (0.149)
  Change at Day 28 | -0.06 (0.185)
  Change at Day 56 | -0.03 (0.057)
  Change at Day 78 | 0.01 (0.098)
  Change at Day 100 | -0.04 (0.075)
  Change at Day 128 | 0.00 (0.063)
  Change at Day 156 | -0.02 (0.053)
  Change at Day 184 | -0.01 (0.079)
  Change at Day 212: number analyzed (Participants) | 6
  Change at Day 212 | 0.04 (0.109)
  Change at Day 240: number analyzed (Participants) | 3
  Change at Day 240 | 0.05 (0.079)
  Change at Day 268: number analyzed (Participants) | 2
  Change at Day 268 | 0.07 (0.096)
  Change at Day 296: number analyzed (Participants) | 2
  Change at Day 296 | 0.04 (0.061)
  Change at Day 324: number analyzed (Participants) | 1
  Change at Day 324 | 0.14 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.

27. Secondary Outcome: Phase 2 (US Population): Change From Baseline in EuroQol Five Dimension Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) Score at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Description: EQ-5D-5L was a 5-item questionnaire consisted of 2 components: a health state profile/a single utility index value and an optional VAS. EQ-5D health state profile/a single utility index value had 5 dimensions including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 5 response levels: 1 =no problems, 2 =slight problems, 3 =moderate problems, 4 =severe problems and 5 =extreme problems. The scores for the 5 dimensions were used to compute a single utility score ranging from 0 to 1 representing the general health status of the individual. Higher score indicated better health status. EQ-5D VAS was used to record participant's rating for his/her "health today" and ranging from 0 to 100, where 0 =worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 53
Score on a scale
  Change at Day 7 | -6.7 [-11.1 to -2.3]
  Change at Day 28 | 0.6 [-3.8 to 5]
  Change at Day 56: number analyzed (Participants) | 51
  Change at Day 56 | 2.2 [-2.3 to 6.7]
  Change at Day 78: number analyzed (Participants) | 46
  Change at Day 78 | 5.3 [0.7 to 9.9]
  Change at Day 100: number analyzed (Participants) | 49
  Change at Day 100 | 1.9 [-2.6 to 6.4]
  Change at Day 128: number analyzed (Participants) | 38
  Change at Day 128 | 6.4 [1.6 to 11.3]
  Change at Day 156: number analyzed (Participants) | 35
  Change at Day 156 | 4.8 [-0.2 to 9.8]
  Change at Day 184: number analyzed (Participants) | 39
  Change at Day 184 | 6.1 [1.2 to 10.9]
  Change at Day 212: number analyzed (Participants) | 33
  Change at Day 212 | 9.6 [4.5 to 14.7]
  Change at Day 240: number analyzed (Participants) | 32
  Change at Day 240 | 11 [5.9 to 16.2]
  Change at Day 268: number analyzed (Participants) | 36
  Change at Day 268 | 7.2 [2.3 to 12.2]
  Change at Day 296: number analyzed (Participants) | 32
  Change at Day 296 | 10 [4.8 to 15.2]
  Change at Day 324: number analyzed (Participants) | 14
  Change at Day 324 | 11.9 [4.9 to 18.9]
  Change at Day 352: number analyzed (Participants) | 7
  Change at Day 352 | 10.2 [0.8 to 19.7]
  Change at Day 380: number analyzed (Participants) | 2
  Change at Day 380 | -2 [-19.1 to 15.1]

28. Secondary Outcome: Phase 2 (Japan Population): Change From Baseline in EuroQol Five Dimension Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) Score at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Description: as for outcome 25
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 8
Score on a scale
  Change at Day 7 | -13.75 (17.269)
  Change at Day 28 | -0.75 (8.795)
  Change at Day 56 | -4.50 (6.803)
  Change at Day 78 | -3.00 (9.914)
  Change at Day 100 | -1.88 (7.530)
  Change at Day 128 | 0.00 (11.019)
  Change at Day 156 | 0.00 (8.452)
  Change at Day 184 | -0.25 (7.005)
  Change at Day 212: number analyzed (Participants) | 6
  Change at Day 212 | 2.50 (9.586)
  Change at Day 240: number analyzed (Participants) | 3
  Change at Day 240 | 0.00 (8.660)
  Change at Day 268: number analyzed (Participants) | 2
  Change at Day 268 | -2.50 (10.607)
  Change at Day 296: number analyzed (Participants) | 2
  Change at Day 296 | -12.50 (24.749)
  Change at Day 324: number analyzed (Participants) | 1
  Change at Day 324 | -10.00 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.

29. Secondary Outcome: Phase 2 (US Population): Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Subscales at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Description: EORTC QLQ-C30 was a 30 items self-reporting questionnaire, with 1 week recall period, resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 Global Health Status scale (GHS), 3 symptom scales (fatigue, nausea and vomiting, and pain) and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Questionnaire includes 28 items with 4-point Likert type responses from "1-not at all" to "4-very much" to assess functioning and symptoms;2 items with 7-point Likert scales (1= poor and 7= excellent) for global health and overall health related QoL. Scores are transformed to 0 to 100 scale, with higher scores representing better GHS, better functioning, and more symptoms. Negative change from baseline values shows deterioration in quality of life or functioning and reduction in symptom and positive values indicate improvement and worsening of symptoms.
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 54
Score on a scale
  Physical functional scales: Change at Day 7 | -14.4 [-19.7 to -9.2]
  Physical functional scales: Change at Day 28: number analyzed (Participants) | 53
  Physical functional scales: Change at Day 28 | -7.2 [-12.4 to -1.9]
  Physical functional scales: Change at Day 56: number analyzed (Participants) | 52
  Physical functional scales: Change at Day 56 | -5.2 [-10.5 to 0.1]
  Physical functional scales: Change at Day 78: number analyzed (Participants) | 47
  Physical functional scales: Change at Day 78 | -2.3 [-7.7 to 3.1]
  Physical functional scales: Change at Day 100: number analyzed (Participants) | 49
  Physical functional scales: Change at Day 100 | -4.8 [-10.2 to 0.5]
  Physical functional scales: Change at Day 128: number analyzed (Participants) | 40
  Physical functional scales: Change at Day 128 | 0 [-5.6 to 5.7]
  Physical functional scales: Change at Day 156: number analyzed (Participants) | 36
  Physical functional scales: Change at Day 156 | -3.9 [-9.7 to 2]
  Physical functional scales: Change at Day 184: number analyzed (Participants) | 40
  Physical functional scales: Change at Day 184 | -0.6 [-6.3 to 5.1]
  Physical functional scales: Change at Day 212: number analyzed (Participants) | 32
  Physical functional scales: Change at Day 212 | 2.2 [-3.9 to 8.2]
  Physical functional scales: Change at Day 240: number analyzed (Participants) | 32
  Physical functional scales: Change at Day 240 | 1.5 [-4.5 to 7.5]
  Physical functional scales: Change at Day 268: number analyzed (Participants) | 36
  Physical functional scales: Change at Day 268 | 2.4 [-3.4 to 8.2]
  Physical functional scales: Change at Day 296: number analyzed (Participants) | 33
  Physical functional scales: Change at Day 296 | 3.1 [-2.9 to 9.1]
  Physical functional scales: Change at Day 324: number analyzed (Participants) | 14
  Physical functional scales: Change at Day 324 | 6.6 [-1.3 to 14.6]
  Physical functional scales: Change at Day 352: number analyzed (Participants) | 7
  Physical functional scales: Change at Day 352 | 6.4 [-4.1 to 16.9]
  Physical functional scales: Change at Day 380: number analyzed (Participants) | 2
  Physical functional scales: Change at Day 380 | -5.5 [-24.2 to 13.2]
  Role functional scales: Change at Day 7 | -24.2 [-32.1 to -16.3]
  Role functional scales: Change at Day 28: number analyzed (Participants) | 53
  Role functional scales: Change at Day 28 | -12.3 [-20.3 to -4.3]
  Role functional scales: Change at Day 56: number analyzed (Participants) | 52
  Role functional scales: Change at Day 56 | -8.5 [-16.5 to -0.4]
  Role functional scales: Change at Day 78: number analyzed (Participants) | 47
  Role functional scales: Change at Day 78 | -3.5 [-11.8 to 4.8]
  Role functional scales: Change at Day 100: number analyzed (Participants) | 49
  Role functional scales: Change at Day 100 | -3 [-11.2 to 5.2]
  Role functional scales: Change at Day 128: number analyzed (Participants) | 40
  Role functional scales: Change at Day 128 | 0.3 [-8.3 to 9]
  Role functional scales: Change at Day 156: number analyzed (Participants) | 36
  Role functional scales: Change at Day 156 | -3.7 [-12.7 to 5.2]
  Role functional scales: Change at Day 184: number analyzed (Participants) | 40
  Role functional scales: Change at Day 184 | 1.1 [-7.6 to 9.7]
  Role functional scales: Change at Day 212: number analyzed (Participants) | 32
  Role functional scales: Change at Day 212 | 0.3 [-8.9 to 9.6]
  Role functional scales: Change at Day 240: number analyzed (Participants) | 32
  Role functional scales: Change at Day 240 | 1.3 [-7.9 to 10.5]
  Role functional scales: Change at Day 268: number analyzed (Participants) | 37
  Role functional scales: Change at Day 268 | 5.5 [-3.4 to 14.3]
  Role functional scales: Change at Day 296: number analyzed (Participants) | 33
  Role functional scales: Change at Day 296 | 4.2 [-5 to 13.3]
  Role functional scales: Change at Day 324: number analyzed (Participants) | 14
  Role functional scales: Change at Day 324 | 7.3 [-5 to 19.6]
  Role functional scales: Change at Day 352: number analyzed (Participants) | 7
  Role functional scales: Change at Day 352 | 8.3 [-8.1 to 24.6]
  Role functional scales: Change at Day 380: number analyzed (Participants) | 2
  Role functional scales: Change at Day 380 | -3.5 [-33 to 25.9]
  Emotional functional scales: Change at Day 7: number analyzed (Participants) | 51
  Emotional functional scales: Change at Day 7 | 3.1 [-1.1 to 7.4]
  Emotional functional scales: Change at Day 28: number analyzed (Participants) | 51
  Emotional functional scales: Change at Day 28 | 6.1 [1.9 to 10.4]
  Emotional functional scales: Change at Day 56: number analyzed (Participants) | 50
  Emotional functional scales: Change at Day 56 | 5.6 [1.3 to 9.9]
  Emotional functional scales: Change at Day 78: number analyzed (Participants) | 45
  Emotional functional scales: Change at Day 78 | 5.7 [1.3 to 10.1]
  Emotional functional scales: Change at Day 100: number analyzed (Participants) | 47
  Emotional functional scales: Change at Day 100 | 4.8 [0.5 to 9.2]
  Emotional functional scales: Change at Day 128: number analyzed (Participants) | 38
  Emotional functional scales: Change at Day 128 | 6.3 [1.7 to 10.9]
  Emotional functional scales: Change at Day 156: number analyzed (Participants) | 35
  Emotional functional scales: Change at Day 156 | 1.7 [-3 to 6.4]
  Emotional functional scales: Change at Day 184: number analyzed (Participants) | 39
  Emotional functional scales: Change at Day 184 | 5.7 [1.1 to 10.3]
  Emotional functional scales: Change at Day 212: number analyzed (Participants) | 33
  Emotional functional scales: Change at Day 212 | 6.3 [1.4 to 11.1]
  Emotional functional scales: Change at Day 240: number analyzed (Participants) | 32
  Emotional functional scales: Change at Day 240 | 7.2 [2.4 to 12.1]
  Emotional functional scales: Change at Day 268: number analyzed (Participants) | 37
  Emotional functional scales: Change at Day 268 | 5.9 [1.3 to 10.6]
  Emotional functional scales: Change at Day 296: number analyzed (Participants) | 33
  Emotional functional scales: Change at Day 296 | 8.4 [3.5 to 13.2]
  Emotional functional scales: Change at Day 324: number analyzed (Participants) | 14
  Emotional functional scales: Change at Day 324 | 12 [5.5 to 18.5]
  Emotional functional scales: Change at Day 352: number analyzed (Participants) | 7
  Emotional functional scales: Change at Day 352 | 8.8 [0.1 to 17.4]
  Emotional functional scales: Change at Day 380: number analyzed (Participants) | 2
  Emotional functional scales: Change at Day 380 | 16 [0.4 to 31.5]
  Cognitive functional scales: Change at Day 7: number analyzed (Participants) | 51
  Cognitive functional scales: Change at Day 7 | -0.4 [-4.8 to 4]
  Cognitive functional scales: Change at Day 28: number analyzed (Participants) | 51
  Cognitive functional scales: Change at Day 28 | 1.6 [-2.8 to 6]
  Cognitive functional scales: Change at Day 56: number analyzed (Participants) | 50
  Cognitive functional scales: Change at Day 56 | 1.2 [-3.3 to 5.6]
  Cognitive functional scales: Change at Day 78: number analyzed (Participants) | 45
  Cognitive functional scales: Change at Day 78 | 4.4 [-0.2 to 9.1]
  Cognitive functional scales: Change at Day 100: number analyzed (Participants) | 47
  Cognitive functional scales: Change at Day 100 | 2.3 [-2.3 to 6.8]
  Cognitive functional scales: Change at Day 128: number analyzed (Participants) | 38
  Cognitive functional scales: Change at Day 128 | 5 [0.1 to 9.9]
  Cognitive functional scales: Change at Day 156: number analyzed (Participants) | 35
  Cognitive functional scales: Change at Day 156 | 4.2 [-0.8 to 9.3]
  Cognitive functional scales: Change at Day 184: number analyzed (Participants) | 39
  Cognitive functional scales: Change at Day 184 | 4.1 [-0.7 to 9]
  Cognitive functional scales: Change at Day 212: number analyzed (Participants) | 33
  Cognitive functional scales: Change at Day 212 | 7.4 [2.2 to 12.5]
  Cognitive functional scales: Change at Day 240: number analyzed (Participants) | 32
  Cognitive functional scales: Change at Day 240 | 8.6 [3.4 to 13.8]
  Cognitive functional scales: Change at Day 268: number analyzed (Participants) | 37
  Cognitive functional scales: Change at Day 268 | 5.6 [0.7 to 10.6]
  Cognitive functional scales: Change at Day 296: number analyzed (Participants) | 33
  Cognitive functional scales: Change at Day 296 | 5.2 [0 to 10.4]
  Cognitive functional scales: Change at Day 324: number analyzed (Participants) | 14
  Cognitive functional scales: Change at Day 324 | 9.3 [2 to 16.6]
  Cognitive functional scales: Change at Day 352: number analyzed (Participants) | 7
  Cognitive functional scales: Change at Day 352 | 4.2 [-5.8 to 14.1]
  Cognitive functional scales: Change at Day 380: number analyzed (Participants) | 2
  Cognitive functional scales: Change at Day 380 | 22 [3.7 to 40.2]
  Social functional scales: Change at Day 7: number analyzed (Participants) | 51
  Social functional scales: Change at Day 7 | -28.5 [-35.6 to -21.5]
  Social functional scales: Change at Day 28: number analyzed (Participants) | 51
  Social functional scales: Change at Day 28 | -13.8 [-20.9 to -6.7]
  Social functional scales: Change at Day 56: number analyzed (Participants) | 50
  Social functional scales: Change at Day 56 | -9.4 [-16.5 to -2.2]
  Social functional scales: Change at Day 78: number analyzed (Participants) | 45
  Social functional scales: Change at Day 78 | -3.8 [-11.2 to 3.6]
  Social functional scales: Change at Day 100: number analyzed (Participants) | 47
  Social functional scales: Change at Day 100 | -3.5 [-10.8 to 3.8]
  Social functional scales: Change at Day 128: number analyzed (Participants) | 38
  Social functional scales: Change at Day 128 | -1.2 [-9 to 6.6]
  Social functional scales: Change at Day 156: number analyzed (Participants) | 35
  Social functional scales: Change at Day 156 | -1.5 [-9.5 to 6.5]
  Social functional scales: Change at Day 184: number analyzed (Participants) | 39
  Social functional scales: Change at Day 184 | 0.4 [-7.4 to 8.1]
  Social functional scales: Change at Day 212: number analyzed (Participants) | 33
  Social functional scales: Change at Day 212 | -1.3 [-9.4 to 6.9]
  Social functional scales: Change at Day 240: number analyzed (Participants) | 32
  Social functional scales: Change at Day 240 | 1.1 [-7.1 to 9.4]
  Social functional scales: Change at Day 268: number analyzed (Participants) | 37
  Social functional scales: Change at Day 268 | -0.5 [-8.3 to 7.4]
  Social functional scales: Change at Day 296: number analyzed (Participants) | 33
  Social functional scales: Change at Day 296 | 2.2 [-5.9 to 10.4]
  Social functional scales: Change at Day 324: number analyzed (Participants) | 14
  Social functional scales: Change at Day 324 | 0.5 [-10.7 to 11.6]
  Social functional scales: Change at Day 352: number analyzed (Participants) | 7
  Social functional scales: Change at Day 352 | -0.1 [-15 to 14.9]
  Social functional scales: Change at Day 380: number analyzed (Participants) | 2
  Social functional scales: Change at Day 380 | -0.5 [-27.7 to 26.6]
  Global health status scale: Change at Day 7: number analyzed (Participants) | 50
  Global health status scale: Change at Day 7 | -9.7 [-15.1 to -4.4]
  Global health status scale: Change at Day 28: number analyzed (Participants) | 51
  Global health status scale: Change at Day 28 | -0.6 [-5.9 to 4.7]
  Global health status scale: Change at Day 56: number analyzed (Participants) | 50
  Global health status scale: Change at Day 56 | 1.5 [-3.9 to 6.8]
  Global health status scale: Change at Day 78: number analyzed (Participants) | 45
  Global health status scale: Change at Day 78 | 4.7 [-0.9 to 10.2]
  Global health status scale: Change at Day 100: number analyzed (Participants) | 47
  Global health status scale: Change at Day 100 | 2.5 [-3 to 8]
  Global health status scale: Change at Day 128: number analyzed (Participants) | 37
  Global health status scale: Change at Day 128 | 8.3 [2.3 to 14.3]
  Global health status scale: Change at Day 156: number analyzed (Participants) | 35
  Global health status scale: Change at Day 156 | 8.4 [2.3 to 14.5]
  Global health status scale: Change at Day 184: number analyzed (Participants) | 39
  Global health status scale: Change at Day 184 | 8.9 [3.1 to 14.8]
  Global health status scale: Change at Day 212: number analyzed (Participants) | 33
  Global health status scale: Change at Day 212 | 7.7 [1.5 to 14]
  Global health status scale: Change at Day 240: number analyzed (Participants) | 32
  Global health status scale: Change at Day 240 | 9.6 [3.3 to 16]
  Global health status scale: Change at Day 268: number analyzed (Participants) | 37
  Global health status scale: Change at Day 268 | 7.8 [1.8 to 13.8]
  Global health status scale: Change at Day 296: number analyzed (Participants) | 33
  Global health status scale: Change at Day 296 | 10.4 [4.2 to 16.7]
  Global health status scale: Change at Day 324: number analyzed (Participants) | 14
  Global health status scale: Change at Day 324 | 11.5 [2.6 to 20.4]
  Global health status scale: Change at Day 352: number analyzed (Participants) | 7
  Global health status scale: Change at Day 352 | 19.9 [7.8 to 32.1]
  Global health status scale: Change at Day 380: number analyzed (Participants) | 2
  Global health status scale: Change at Day 380 | 4.4 [-17.9 to 26.8]
  Pain symptom scales: Change at Day 7 | -1.9 [-8.5 to 4.6]
  Pain symptom scales: Change at Day 28: number analyzed (Participants) | 53
  Pain symptom scales: Change at Day 28 | -9.9 [-16.5 to -3.3]
  Pain symptom scales: Change at Day 56: number analyzed (Participants) | 52
  Pain symptom scales: Change at Day 56 | -6.3 [-12.9 to 0.4]
  Pain symptom scales: Change at Day 78: number analyzed (Participants) | 47
  Pain symptom scales: Change at Day 78 | -9.4 [-16.3 to -2.5]
  Pain symptom scales: Change at Day 100: number analyzed (Participants) | 50
  Pain symptom scales: Change at Day 100 | -10.5 [-17.3 to -3.8]
  Pain symptom scales: Change at Day 128: number analyzed (Participants) | 40
  Pain symptom scales: Change at Day 128 | -11.8 [-19.1 to -4.6]
  Pain symptom scales: Change at Day 156: number analyzed (Participants) | 36
  Pain symptom scales: Change at Day 156 | -13.1 [-20.6 to -5.5]
  Pain symptom scales: Change at Day 184: number analyzed (Participants) | 40
  Pain symptom scales: Change at Day 184 | -10 [-17.3 to -2.7]
  Pain symptom scales: Change at Day 212: number analyzed (Participants) | 33
  Pain symptom scales: Change at Day 212 | -11.7 [-19.5 to -3.9]
  Pain symptom scales: Change at Day 240: number analyzed (Participants) | 32
  Pain symptom scales: Change at Day 240 | -16.2 [-24.1 to -8.3]
  Pain symptom scales: Change at Day 268: number analyzed (Participants) | 37
  Pain symptom scales: Change at Day 268 | -16.7 [-24.2 to -9.2]
  Pain symptom scales: Change at Day 296: number analyzed (Participants) | 33
  Pain symptom scales: Change at Day 296 | -15.6 [-23.5 to -7.8]
  Pain symptom scales: Change at Day 324: number analyzed (Participants) | 14
  Pain symptom scales: Change at Day 324 | -14.9 [-25.9 to -3.9]
  Pain symptom scales: Change at Day 352: number analyzed (Participants) | 7
  Pain symptom scales: Change at Day 352 | -17.6 [-32.6 to -2.6]
  Pain symptom scales: Change at Day 380: number analyzed (Participants) | 2
  Pain symptom scales: Change at Day 380 | -0.7 [-28.2 to 26.7]
  Fatigue symptom scales: Change at Day 7 | 14.3 [8.7 to 20]
  Fatigue symptom scales: Change at Day 28: number analyzed (Participants) | 53
  Fatigue symptom scales: Change at Day 28 | 10.3 [4.6 to 16.1]
  Fatigue symptom scales: Change at Day 56: number analyzed (Participants) | 52
  Fatigue symptom scales: Change at Day 56 | 4 [-1.7 to 9.7]
  Fatigue symptom scales: Change at Day 78: number analyzed (Participants) | 47
  Fatigue symptom scales: Change at Day 78 | -5.9 [-11.8 to 0]
  Fatigue symptom scales: Change at Day 100: number analyzed (Participants) | 49
  Fatigue symptom scales: Change at Day 100 | 0 [-5.9 to 5.8]
  Fatigue symptom scales: Change at Day 128: number analyzed (Participants) | 40
  Fatigue symptom scales: Change at Day 128 | -7.7 [-13.9 to -1.5]
  Fatigue symptom scales: Change at Day 156: number analyzed (Participants) | 36
  Fatigue symptom scales: Change at Day 156 | -5.1 [-11.5 to 1.2]
  Fatigue symptom scales: Change at Day 184: number analyzed (Participants) | 40
  Fatigue symptom scales: Change at Day 184 | -8.1 [-14.3 to -1.9]
  Fatigue symptom scales: Change at Day 212: number analyzed (Participants) | 32
  Fatigue symptom scales: Change at Day 212 | -11.5 [-18.1 to -4.8]
  Fatigue symptom scales: Change at Day 240: number analyzed (Participants) | 32
  Fatigue symptom scales: Change at Day 240 | -12.6 [-19.2 to -5.9]
  Fatigue symptom scales: Change at Day 268: number analyzed (Participants) | 37
  Fatigue symptom scales: Change at Day 268 | -13.4 [-19.8 to -7.1]
  Fatigue symptom scales: Change at Day 296: number analyzed (Participants) | 33
  Fatigue symptom scales: Change at Day 296 | -14.2 [-20.8 to -7.6]
  Fatigue symptom scales: Change at Day 324: number analyzed (Participants) | 14
  Fatigue symptom scales: Change at Day 324 | -14.6 [-23.6 to -5.6]
  Fatigue symptom scales: Change at Day 352: number analyzed (Participants) | 7
  Fatigue symptom scales: Change at Day 352 | -15.7 [-27.7 to -3.7]
  Fatigue symptom scales: Change at Day 380: number analyzed (Participants) | 2
  Fatigue symptom scales: Change at Day 380 | -5.6 [-27.3 to 16.1]
  Nausea/vomiting symptom scales: Change at Day 7 | 13.3 [9.8 to 16.9]
  Nausea/vomiting symptom scales: Change at Day 28: number analyzed (Participants) | 53
  Nausea/vomiting symptom scales: Change at Day 28 | 1.7 [-1.9 to 5.3]
  Nausea/vomiting symptom scales: Change at Day 56: number analyzed (Participants) | 52
  Nausea/vomiting symptom scales: Change at Day 56 | 2.2 [-1.5 to 5.8]
  Nausea/vomiting symptom scales: Change at Day 78: number analyzed (Participants) | 47
  Nausea/vomiting symptom scales: Change at Day 78 | -0.2 [-4 to 3.6]
  Nausea/vomiting symptom scales: Change at Day 100: number analyzed (Participants) | 49
  Nausea/vomiting symptom scales: Change at Day 100 | -0.2 [-4 to 3.5]
  Nausea/vomiting symptom scales: Change at Day 128: number analyzed (Participants) | 40
  Nausea/vomiting symptom scales: Change at Day 128 | -2.6 [-6.6 to 1.5]
  Nausea/vomiting symptom scales: Change at Day 156: number analyzed (Participants) | 36
  Nausea/vomiting symptom scales: Change at Day 156 | -2.6 [-6.9 to 1.6]
  Nausea/vomiting symptom scales: Change at Day 184: number analyzed (Participants) | 40
  Nausea/vomiting symptom scales: Change at Day 184 | -0.2 [-4.2 to 3.9]
  Nausea/vomiting symptom scales: Change at Day 212: number analyzed (Participants) | 32
  Nausea/vomiting symptom scales: Change at Day 212 | -1 [-5.5 to 3.5]
  Nausea/vomiting symptom scales: Change at Day 240: number analyzed (Participants) | 32
  Nausea/vomiting symptom scales: Change at Day 240 | -3.4 [-7.9 to 1]
  Nausea/vomiting symptom scales: Change at Day 268: number analyzed (Participants) | 37
  Nausea/vomiting symptom scales: Change at Day 268 | -2.5 [-6.7 to 1.7]
  Nausea/vomiting symptom scales: Change at Day 296: number analyzed (Participants) | 33
  Nausea/vomiting symptom scales: Change at Day 296 | -3.5 [-7.9 to 1]
  Nausea/vomiting symptom scales: Change at Day 324: number analyzed (Participants) | 14
  Nausea/vomiting symptom scales: Change at Day 324 | -2.9 [-9.4 to 3.6]
  Nausea/vomiting symptom scales: Change at Day 352: number analyzed (Participants) | 7
  Nausea/vomiting symptom scales: Change at Day 352 | -4.4 [-13.4 to 4.6]
  Nausea/vomiting symptom scales: Change at Day 380: number analyzed (Participants) | 2
  Nausea/vomiting symptom scales: Change at Day 380 | 4.5 [-12.3 to 21.2]
  Dyspnea: Change at Day 7 | 2.6 [-2.7 to 8]
  Dyspnea: Change at Day 28: number analyzed (Participants) | 53
  Dyspnea: Change at Day 28 | 4.6 [-0.8 to 10]
  Dyspnea: Change at Day 56: number analyzed (Participants) | 52
  Dyspnea: Change at Day 56 | 1.3 [-4.1 to 6.8]
  Dyspnea: Change at Day 78: number analyzed (Participants) | 47
  Dyspnea: Change at Day 78 | -1.9 [-7.6 to 3.8]
  Dyspnea: Change at Day 100: number analyzed (Participants) | 48
  Dyspnea: Change at Day 100 | -3 [-8.7 to 2.6]
  Dyspnea: Change at Day 128: number analyzed (Participants) | 39
  Dyspnea: Change at Day 128 | -1.5 [-7.6 to 4.6]
  Dyspnea: Change at Day 156: number analyzed (Participants) | 36
  Dyspnea: Change at Day 156 | -1.3 [-7.6 to 5]
  Dyspnea: Change at Day 184: number analyzed (Participants) | 40
  Dyspnea: Change at Day 184 | -2.9 [-8.9 to 3.2]
  Dyspnea: Change at Day 212: number analyzed (Participants) | 32
  Dyspnea: Change at Day 212 | -7 [-13.6 to -0.4]
  Dyspnea: Change at Day 240: number analyzed (Participants) | 32
  Dyspnea: Change at Day 240 | -4.1 [-10.7 to 2.5]
  Dyspnea: Change at Day 268: number analyzed (Participants) | 37
  Dyspnea: Change at Day 268 | -8.7 [-15 to -2.5]
  Dyspnea: Change at Day 296: number analyzed (Participants) | 33
  Dyspnea: Change at Day 296 | -10.9 [-17.5 to -4.4]
  Dyspnea: Change at Day 324: number analyzed (Participants) | 14
  Dyspnea: Change at Day 324 | -7.6 [-17 to 1.8]
  Dyspnea: Change at Day 352: number analyzed (Participants) | 7
  Dyspnea: Change at Day 352 | -6.5 [-19.4 to 6.4]
  Dyspnea: Change at Day 380: number analyzed (Participants) | 2
  Dyspnea: Change at Day 380 | -22.5 [-46.3 to 1.4]
  Insomnia: Change at Day 7 | 9.4 [2.9 to 15.9]
  Insomnia: Change at Day 28: number analyzed (Participants) | 52
  Insomnia: Change at Day 28 | -4.6 [-11.2 to 2]
  Insomnia: Change at Day 56: number analyzed (Participants) | 52
  Insomnia: Change at Day 56 | -1.4 [-8 to 5.3]
  Insomnia: Change at Day 78: number analyzed (Participants) | 47
  Insomnia: Change at Day 78 | -2.6 [-9.5 to 4.3]
  Insomnia: Change at Day 100: number analyzed (Participants) | 49
  Insomnia: Change at Day 100 | -3.1 [-9.9 to 3.6]
  Insomnia: Change at Day 128: number analyzed (Participants) | 40
  Insomnia: Change at Day 128 | -7.1 [-14.4 to 0.2]
  Insomnia: Change at Day 156: number analyzed (Participants) | 36
  Insomnia: Change at Day 156 | -7.1 [-14.7 to 0.5]
  Insomnia: Change at Day 184: number analyzed (Participants) | 40
  Insomnia: Change at Day 184 | -2.3 [-9.6 to 5]
  Insomnia: Change at Day 212: number analyzed (Participants) | 32
  Insomnia: Change at Day 212 | -4.4 [-12.4 to 3.5]
  Insomnia: Change at Day 240: number analyzed (Participants) | 32
  Insomnia: Change at Day 240 | -6.3 [-14.2 to 1.7]
  Insomnia: Change at Day 268: number analyzed (Participants) | 37
  Insomnia: Change at Day 268 | -6.7 [-14.3 to 0.8]
  Insomnia: Change at Day 296: number analyzed (Participants) | 33
  Insomnia: Change at Day 296 | -4.9 [-12.8 to 3]
  Insomnia: Change at Day 324: number analyzed (Participants) | 14
  Insomnia: Change at Day 324 | -1.6 [-12.9 to 9.6]
  Insomnia: Change at Day 352: number analyzed (Participants) | 7
  Insomnia: Change at Day 352 | 1 [-14.4 to 16.5]
  Insomnia: Change at Day 380: number analyzed (Participants) | 2
  Insomnia: Change at Day 380 | -18.3 [-46.7 to 10.1]
  Appetite loss: Change at Day 7 | 22.2 [16 to 28.4]
  Appetite loss: Change at Day 28: number analyzed (Participants) | 53
  Appetite loss: Change at Day 28 | 8.4 [2.1 to 14.6]
  Appetite loss: Change at Day 56: number analyzed (Participants) | 52
  Appetite loss: Change at Day 56 | 2.5 [-3.8 to 8.8]
  Appetite loss: Change at Day 78: number analyzed (Participants) | 47
  Appetite loss: Change at Day 78 | -0.7 [-7.3 to 5.8]
  Appetite loss: Change at Day 100: number analyzed (Participants) | 49
  Appetite loss: Change at Day 100 | 3 [-3.5 to 9.4]
  Appetite loss: Change at Day 128: number analyzed (Participants) | 40
  Appetite loss: Change at Day 128 | -4.3 [-11.3 to 2.7]
  Appetite loss: Change at Day 156: number analyzed (Participants) | 36
  Appetite loss: Change at Day 156 | -5 [-12.3 to 2.3]
  Appetite loss: Change at Day 184: number analyzed (Participants) | 40
  Appetite loss: Change at Day 184 | -4.7 [-11.7 to 2.2]
  Appetite loss: Change at Day 212: number analyzed (Participants) | 32
  Appetite loss: Change at Day 212 | -7.9 [-15.5 to -0.3]
  Appetite loss: Change at Day 240: number analyzed (Participants) | 32
  Appetite loss: Change at Day 240 | -10.5 [-18.1 to -2.9]
  Appetite loss: Change at Day 268: number analyzed (Participants) | 37
  Appetite loss: Change at Day 268 | -12.4 [-19.6 to -5.2]
  Appetite loss: Change at Day 296: number analyzed (Participants) | 33
  Appetite loss: Change at Day 296 | -11 [-18.5 to -3.4]
  Appetite loss: Change at Day 324: number analyzed (Participants) | 14
  Appetite loss: Change at Day 324 | -9.5 [-20.4 to 1.3]
  Appetite loss: Change at Day 352: number analyzed (Participants) | 7
  Appetite loss: Change at Day 352 | -9.8 [-24.8 to 5.2]
  Appetite loss: Change at Day 380: number analyzed (Participants) | 2
  Appetite loss: Change at Day 380 | -6.1 [-33.7 to 21.5]
  Constipation: Change at Day 7 | 12.7 [8.4 to 17]
  Constipation: Change at Day 28: number analyzed (Participants) | 53
  Constipation: Change at Day 28 | -0.1 [-4.5 to 4.2]
  Constipation: Change at Day 56: number analyzed (Participants) | 52
  Constipation: Change at Day 56 | -2 [-6.4 to 2.4]
  Constipation: Change at Day 78: number analyzed (Participants) | 47
  Constipation: Change at Day 78 | -6.3 [-10.9 to -1.7]
  Constipation: Change at Day 100: number analyzed (Participants) | 49
  Constipation: Change at Day 100 | -7 [-11.5 to -2.5]
  Constipation: Change at Day 128: number analyzed (Participants) | 40
  Constipation: Change at Day 128 | -4.5 [-9.4 to 0.5]
  Constipation: Change at Day 156: number analyzed (Participants) | 36
  Constipation: Change at Day 156 | -6.3 [-11.5 to -1.2]
  Constipation: Change at Day 184: number analyzed (Participants) | 40
  Constipation: Change at Day 184 | -8.1 [-13 to -3.2]
  Constipation: Change at Day 212: number analyzed (Participants) | 32
  Constipation: Change at Day 212 | -4.4 [-9.8 to 1.1]
  Constipation: Change at Day 240: number analyzed (Participants) | 32
  Constipation: Change at Day 240 | -10.1 [-15.5 to -4.6]
  Constipation: Change at Day 268: number analyzed (Participants) | 37
  Constipation: Change at Day 268 | -6.6 [-11.7 to -1.5]
  Constipation: Change at Day 296: number analyzed (Participants) | 33
  Constipation: Change at Day 296 | -7.1 [-12.4 to -1.7]
  Constipation: Change at Day 324: number analyzed (Participants) | 14
  Constipation: Change at Day 324 | -9.3 [-17.2 to -1.4]
  Constipation: Change at Day 352: number analyzed (Participants) | 7
  Constipation: Change at Day 352 | -12.3 [-23.3 to -1.3]
  Constipation: Change at Day 380: number analyzed (Participants) | 2
  Constipation: Change at Day 380 | -16.5 [-36 to 36.9]
  Diarrhea: Change at Day 7: number analyzed (Participants) | 51
  Diarrhea: Change at Day 7 | 1.7 [-3.6 to 6.9]
  Diarrhea: Change at Day 28: number analyzed (Participants) | 50
  Diarrhea: Change at Day 28 | -3.1 [-8.4 to 2.2]
  Diarrhea: Change at Day 56: number analyzed (Participants) | 50
  Diarrhea: Change at Day 56 | 1.2 [-4.1 to 6.5]
  Diarrhea: Change at Day 78: number analyzed (Participants) | 45
  Diarrhea: Change at Day 78 | 5 [-0.5 to 10.6]
  Diarrhea: Change at Day 100: number analyzed (Participants) | 47
  Diarrhea: Change at Day 100 | 0.1 [-5.3 to 5.5]
  Diarrhea: Change at Day 128: number analyzed (Participants) | 38
  Diarrhea: Change at Day 128 | -1.6 [-7.5 to 4.3]
  Diarrhea: Change at Day 156: number analyzed (Participants) | 35
  Diarrhea: Change at Day 156 | 1.1 [-5 to 7.2]
  Diarrhea: Change at Day 184: number analyzed (Participants) | 39
  Diarrhea: Change at Day 184 | -4.5 [-10.3 to 1.4]
  Diarrhea: Change at Day 212: number analyzed (Participants) | 33
  Diarrhea: Change at Day 212 | -6.8 [-13.1 to -0.6]
  Diarrhea: Change at Day 240: number analyzed (Participants) | 32
  Diarrhea: Change at Day 240 | -2.6 [-9 to 3.7]
  Diarrhea: Change at Day 268: number analyzed (Participants) | 37
  Diarrhea: Change at Day 268 | -5.4 [-11.3 to 0.6]
  Diarrhea: Change at Day 296: number analyzed (Participants) | 33
  Diarrhea: Change at Day 296 | -8.2 [-14.5 to -2]
  Diarrhea: Change at Day 324: number analyzed (Participants) | 14
  Diarrhea: Change at Day 324 | -12.2 [-21.3 to -3]
  Diarrhea: Change at Day 352: number analyzed (Participants) | 7
  Diarrhea: Change at Day 352 | -11.9 [-24.5 to 0.7]
  Diarrhea: Change at Day 380: number analyzed (Participants) | 2
  Diarrhea: Change at Day 380 | -26.2 [-49.5 to -2.9]
  Financial difficulties: Change at Day 7: number analyzed (Participants) | 50
  Financial difficulties: Change at Day 7 | 3.8 [-2.5 to 10]
  Financial difficulties: Change at Day 28: number analyzed (Participants) | 51
  Financial difficulties: Change at Day 28 | -2.7 [-8.9 to 3.6]
  Financial difficulties: Change at Day 56: number analyzed (Participants) | 49
  Financial difficulties: Change at Day 56 | -1.4 [-7.7 to 4.9]
  Financial difficulties: Change at Day 78: number analyzed (Participants) | 45
  Financial difficulties: Change at Day 78 | -4.5 [-10.9 to 2]
  Financial difficulties: Change at Day 100: number analyzed (Participants) | 47
  Financial difficulties: Change at Day 100 | -4.3 [-10.7 to 2.1]
  Financial difficulties: Change at Day 128: number analyzed (Participants) | 38
  Financial difficulties: Change at Day 128 | -6.4 [-13.3 to 0.4]
  Financial difficulties: Change at Day 156: number analyzed (Participants) | 35
  Financial difficulties: Change at Day 156 | -4.7 [-11.7 to 2.3]
  Financial difficulties: Change at Day 184: number analyzed (Participants) | 39
  Financial difficulties: Change at Day 184 | -5.2 [-11.9 to 1.6]
  Financial difficulties: Change at Day 212: number analyzed (Participants) | 33
  Financial difficulties: Change at Day 212 | -2.7 [-9.8 to 4.4]
  Financial difficulties: Change at Day 240: number analyzed (Participants) | 32
  Financial difficulties: Change at Day 240 | -4.1 [-11.3 to 3.1]
  Financial difficulties: Change at Day 268: number analyzed (Participants) | 37
  Financial difficulties: Change at Day 268 | -9.1 [-15.9 to -2.2]
  Financial difficulties: Change at Day 296: number analyzed (Participants) | 33
  Financial difficulties: Change at Day 296 | -8.3 [-15.5 to -1.2]
  Financial difficulties: Change at Day 324: number analyzed (Participants) | 14
  Financial difficulties: Change at Day 324 | -12 [-21.7 to -2.3]
  Financial difficulties: Change at Day 352: number analyzed (Participants) | 7
  Financial difficulties: Change at Day 352 | -12.8 [-25.8 to 0.2]
  Financial difficulties: Change at Day 380: number analyzed (Participants) | 2
  Financial difficulties: Change at Day 380 | -21.2 [-44.6 to 2.3]

30. Secondary Outcome: Phase 2 (Japan Population): Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Subscales at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Description: as for outcome 29
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 8
Score on a scale
  Physical functional scales: Change at Day 7 | -2.50 (12.312)
  Physical functional scales: Change at Day 28 | -4.17 (10.040)
  Physical functional scales: Change at Day 56 | -1.67 (6.901)
  Physical functional scales: Change at Day 78 | 0.00 (3.563)
  Physical functional scales: Change at Day 100 | -1.67 (5.909)
  Physical functional scales: Change at Day 128 | -0.83 (8.309)
  Physical functional scales: Change at Day 156 | 0.83 (6.607)
  Physical functional scales: Change at Day 184 | 4.17 (4.960)
  Physical functional scales: Change at Day 212: number analyzed (Participants) | 6
  Physical functional scales: Change at Day 212 | 4.44 (5.443)
  Physical functional scales: Change at Day 240: number analyzed (Participants) | 3
  Physical functional scales: Change at Day 240 | 4.44 (7.698)
  Physical functional scales: Change at Day 268: number analyzed (Participants) | 2
  Physical functional scales: Change at Day 268 | -3.33 (4.714)
  Physical functional scales: Change at Day 296: number analyzed (Participants) | 2
  Physical functional scales: Change at Day 296 | 0.00 (0.000)
  Physical functional scales: Change at Day 324: number analyzed (Participants) | 1
  Physical functional scales: Change at Day 324 | 0.00
  Role functional scales: Change at Day 7 | -10.42 (15.269)
  Role functional scales: Change at Day 28 | -8.33 (17.817)
  Role functional scales: Change at Day 56 | -12.50 (17.252)
  Role functional scales: Change at Day 78 | -6.25 (26.633)
  Role functional scales: Change at Day 100 | -6.25 (15.269)
  Role functional scales: Change at Day 128 | -16.67 (26.726)
  Role functional scales: Change at Day 156 | -10.42 (26.633)
  Role functional scales: Change at Day 184 | -10.42 (29.463)
  Role functional scales: Change at Day 212: number analyzed (Participants) | 6
  Role functional scales: Change at Day 212 | -8.33 (20.412)
  Role functional scales: Change at Day 240: number analyzed (Participants) | 3
  Role functional scales: Change at Day 240 | -11.11 (19.245)
  Role functional scales: Change at Day 268: number analyzed (Participants) | 2
  Role functional scales: Change at Day 268 | -8.33 (11.785)
  Role functional scales: Change at Day 296: number analyzed (Participants) | 2
  Role functional scales: Change at Day 296 | -16.67 (23.570)
  Role functional scales: Change at Day 324: number analyzed (Participants) | 1
  Role functional scales: Change at Day 324 | -16.67 (NA) — Standard deviation (SD) could not be calculated as only 1 participant was available.
  Emotional functional scales: Change at Day 7 | 2.08 (9.708)
  Emotional functional scales: Change at Day 28 | 1.04 (8.259)
  Emotional functional scales: Change at Day 56 | 6.25 (8.626)
  Emotional functional scales: Change at Day 78 | 4.17 (9.960)
  Emotional functional scales: Change at Day 100 | 5.21 (8.839)
  Emotional functional scales: Change at Day 128 | 3.13 (11.732)
  Emotional functional scales: Change at Day 156 | 5.21 (9.898)
  Emotional functional scales: Change at Day 184 | 9.38 (6.954)
  Emotional functional scales: Change at Day 212: number analyzed (Participants) | 6
  Emotional functional scales: Change at Day 212 | 2.78 (6.804)
  Emotional functional scales: Change at Day 240: number analyzed (Participants) | 3
  Emotional functional scales: Change at Day 240 | 11.11 (9.623)
  Emotional functional scales: Change at Day 268: number analyzed (Participants) | 2
  Emotional functional scales: Change at Day 268 | 8.33 (11.785)
  Emotional functional scales: Change at Day 296: number analyzed (Participants) | 2
  Emotional functional scales: Change at Day 296 | -4.17 (5.893)
  Emotional functional scales: Change at Day 324: number analyzed (Participants) | 1
  Emotional functional scales: Change at Day 324 | 16.67 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Cognitive functional scales: Change at Day 7 | -4.17 (11.785)
  Cognitive functional scales: Change at Day 28 | 2.08 (5.893)
  Cognitive functional scales: Change at Day 56 | -4.17 (14.773)
  Cognitive functional scales: Change at Day 78 | 0.00 (12.599)
  Cognitive functional scales: Change at Day 100 | -2.08 (10.681)
  Cognitive functional scales: Change at Day 128 | -4.17 (11.785)
  Cognitive functional scales: Change at Day 156 | 0.00 (15.430)
  Cognitive functional scales: Change at Day 184 | 2.08 (13.909)
  Cognitive functional scales: Change at Day 212: number analyzed (Participants) | 6
  Cognitive functional scales: Change at Day 212 | 0.00 (14.907)
  Cognitive functional scales: Change at Day 240: number analyzed (Participants) | 3
  Cognitive functional scales: Change at Day 240 | 11.11 (9.623)
  Cognitive functional scales: Change at Day 268: number analyzed (Participants) | 2
  Cognitive functional scales: Change at Day 268 | 8.33 (11.785)
  Cognitive functional scales: Change at Day 296: number analyzed (Participants) | 2
  Cognitive functional scales: Change at Day 296 | -8.33 (11.785)
  Cognitive functional scales: Change at Day 324: number analyzed (Participants) | 1
  Cognitive functional scales: Change at Day 324 | 0.00 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Social functional scales: Change at Day 7 | -2.08 (20.774)
  Social functional scales: Change at Day 28 | 2.08 (5.893)
  Social functional scales: Change at Day 56 | 4.17 (7.715)
  Social functional scales: Change at Day 78 | -2.08 (16.517)
  Social functional scales: Change at Day 100 | 4.17 (19.416)
  Social functional scales: Change at Day 128 | 0.00 (8.909)
  Social functional scales: Change at Day 156 | 0.00 (15.430)
  Social functional scales: Change at Day 184 | 6.25 (12.400)
  Social functional scales: Change at Day 212: number analyzed (Participants) | 6
  Social functional scales: Change at Day 212 | 0.00 (10.541)
  Social functional scales: Change at Day 240: number analyzed (Participants) | 3
  Social functional scales: Change at Day 240 | 11.11 (9.623)
  Social functional scales: Change at Day 268: number analyzed (Participants) | 2
  Social functional scales: Change at Day 268 | 16.67 (23.570)
  Social functional scales: Change at Day 296: number analyzed (Participants) | 2
  Social functional scales: Change at Day 296 | 0.00 (0.000)
  Social functional scales: Change at Day 324: number analyzed (Participants) | 1
  Social functional scales: Change at Day 324 | 33.33 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Global health status scale: Change at Day 7 | -8.33 (15.430)
  Global health status scale: Change at Day 28 | -13.54 (30.190)
  Global health status scale: Change at Day 56 | -4.17 (17.817)
  Global health status scale: Change at Day 78 | -6.25 (8.626)
  Global health status scale: Change at Day 100 | -2.08 (13.176)
  Global health status scale: Change at Day 128 | -3.13 (17.783)
  Global health status scale: Change at Day 156 | -3.13 (14.042)
  Global health status scale: Change at Day 184 | -5.21 (13.317)
  Global health status scale: Change at Day 212: number analyzed (Participants) | 6
  Global health status scale: Change at Day 212 | -2.78 (6.804)
  Global health status scale: Change at Day 240: number analyzed (Participants) | 3
  Global health status scale: Change at Day 240 | 5.56 (12.729)
  Global health status scale: Change at Day 268: number analyzed (Participants) | 2
  Global health status scale: Change at Day 268 | 12.50 (5.893)
  Global health status scale: Change at Day 296: number analyzed (Participants) | 2
  Global health status scale: Change at Day 296 | -4.17 (17.678)
  Global health status scale: Change at Day 324: number analyzed (Participants) | 1
  Global health status scale: Change at Day 324 | 16.67 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Pain symptom scales: Change at Day 7 | 20.83 (30.538)
  Pain symptom scales: Change at Day 28 | -2.08 (10.681)
  Pain symptom scales: Change at Day 56 | 8.33 (17.817)
  Pain symptom scales: Change at Day 78 | 4.17 (14.773)
  Pain symptom scales: Change at Day 100 | 2.08 (10.681)
  Pain symptom scales: Change at Day 128 | 4.17 (19.416)
  Pain symptom scales: Change at Day 156 | 0.00 (12.599)
  Pain symptom scales: Change at Day 184 | 2.08 (5.893)
  Pain symptom scales: Change at Day 212: number analyzed (Participants) | 6
  Pain symptom scales: Change at Day 212 | -2.78 (12.546)
  Pain symptom scales: Change at Day 240: number analyzed (Participants) | 3
  Pain symptom scales: Change at Day 240 | -5.56 (9.623)
  Pain symptom scales: Change at Day 268: number analyzed (Participants) | 2
  Pain symptom scales: Change at Day 268 | -8.33 (11.785)
  Pain symptom scales: Change at Day 296: number analyzed (Participants) | 2
  Pain symptom scales: Change at Day 296 | 0.00 (23.570)
  Pain symptom scales: Change at Day 324: number analyzed (Participants) | 1
  Pain symptom scales: Change at Day 324 | 0.00 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Fatigue symptom scales: Change at Day 7 | 4.17 (30.825)
  Fatigue symptom scales: Change at Day 28 | 1.39 (13.849)
  Fatigue symptom scales: Change at Day 56 | 6.94 (10.179)
  Fatigue symptom scales: Change at Day 78 | 6.94 (13.197)
  Fatigue symptom scales: Change at Day 100 | 2.78 (9.849)
  Fatigue symptom scales: Change at Day 128 | 6.94 (19.642)
  Fatigue symptom scales: Change at Day 156 | 2.78 (7.857)
  Fatigue symptom scales: Change at Day 184 | 0.00 (5.939)
  Fatigue symptom scales: Change at Day 212: number analyzed (Participants) | 6
  Fatigue symptom scales: Change at Day 212 | -5.56 (9.296)
  Fatigue symptom scales: Change at Day 240: number analyzed (Participants) | 3
  Fatigue symptom scales: Change at Day 240 | 3.70 (35.717)
  Fatigue symptom scales: Change at Day 268: number analyzed (Participants) | 2
  Fatigue symptom scales: Change at Day 268 | 0.00 (15.713)
  Fatigue symptom scales: Change at Day 296: number analyzed (Participants) | 2
  Fatigue symptom scales: Change at Day 296 | 16.67 (23.570)
  Fatigue symptom scales: Change at Day 324: number analyzed (Participants) | 1
  Fatigue symptom scales: Change at Day 324 | 11.11 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Nausea/vomiting symptom scales: Change at Day 7 | 14.58 (18.767)
  Nausea/vomiting symptom scales: Change at Day 28 | 2.08 (5.893)
  Nausea/vomiting symptom scales: Change at Day 56 | 2.08 (5.893)
  Nausea/vomiting symptom scales: Change at Day 78 | 2.08 (5.893)
  Nausea/vomiting symptom scales: Change at Day 100 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 128 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 156 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 184 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 212: number analyzed (Participants) | 6
  Nausea/vomiting symptom scales: Change at Day 212 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 240: number analyzed (Participants) | 3
  Nausea/vomiting symptom scales: Change at Day 240 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 268: number analyzed (Participants) | 2
  Nausea/vomiting symptom scales: Change at Day 268 | 0.00 (0.000)
  Nausea/vomiting symptom scales: Change at Day 296: number analyzed (Participants) | 2
  Nausea/vomiting symptom scales: Change at Day 296 | 0.00 (47.140)
  Nausea/vomiting symptom scales: Change at Day 324: number analyzed (Participants) | 1
  Nausea/vomiting symptom scales: Change at Day 324 | 0.00 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Dyspnea: Change at Day 7 | 4.17 (45.207)
  Dyspnea: Change at Day 28 | -12.50 (24.801)
  Dyspnea: Change at Day 56 | -4.17 (21.362)
  Dyspnea: Change at Day 78 | 8.33 (29.547)
  Dyspnea: Change at Day 100 | 0.00 (17.817)
  Dyspnea: Change at Day 128 | -8.33 (15.430)
  Dyspnea: Change at Day 156 | -12.50 (24.801)
  Dyspnea: Change at Day 184 | -12.50 (24.801)
  Dyspnea: Change at Day 212: number analyzed (Participants) | 6
  Dyspnea: Change at Day 212 | -16.67 (27.889)
  Dyspnea: Change at Day 240: number analyzed (Participants) | 3
  Dyspnea: Change at Day 240 | -11.11 (38.490)
  Dyspnea: Change at Day 268: number analyzed (Participants) | 2
  Dyspnea: Change at Day 268 | 0.00 (47.140)
  Dyspnea: Change at Day 296: number analyzed (Participants) | 2
  Dyspnea: Change at Day 296 | 0.00 (47.140)
  Dyspnea: Change at Day 324: number analyzed (Participants) | 1
  Dyspnea: Change at Day 324 | 33.33 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Insomnia: Change at Day 7 | 8.33 (23.570)
  Insomnia: Change at Day 28 | -4.17 (21.362)
  Insomnia: Change at Day 56 | -4.17 (21.362)
  Insomnia: Change at Day 78 | 0.00 (17.817)
  Insomnia: Change at Day 100 | 4.17 (11.785)
  Insomnia: Change at Day 128 | -4.17 (21.362)
  Insomnia: Change at Day 156 | -4.17 (21.362)
  Insomnia: Change at Day 184 | -8.33 (15.430)
  Insomnia: Change at Day 212: number analyzed (Participants) | 6
  Insomnia: Change at Day 212 | 0.00 (21.082)
  Insomnia: Change at Day 240: number analyzed (Participants) | 3
  Insomnia: Change at Day 240 | -11.11 (19.245)
  Insomnia: Change at Day 268: number analyzed (Participants) | 2
  Insomnia: Change at Day 268 | -16.67 (23.570)
  Insomnia: Change at Day 296: number analyzed (Participants) | 2
  Insomnia: Change at Day 296 | 16.67 (23.570)
  Insomnia: Change at Day 324: number analyzed (Participants) | 1
  Insomnia: Change at Day 324 | 0.00
  Appetite loss: Change at Day 7 | 20.83 (24.801)
  Appetite loss: Change at Day 28 | 16.67 (17.817)
  Appetite loss: Change at Day 56 | 4.17 (11.785)
  Appetite loss: Change at Day 78 | 8.33 (15.430)
  Appetite loss: Change at Day 100 | 4.17 (11.785)
  Appetite loss: Change at Day 128 | 16.67 (25.198)
  Appetite loss: Change at Day 156 | 4.17 (11.785)
  Appetite loss: Change at Day 184 | 4.17 (11.785)
  Appetite loss: Change at Day 212: number analyzed (Participants) | 6
  Appetite loss: Change at Day 212 | 0.00 (0.000)
  Appetite loss: Change at Day 240: number analyzed (Participants) | 3
  Appetite loss: Change at Day 240 | 0.00 (0.000)
  Appetite loss: Change at Day 268: number analyzed (Participants) | 3
  Appetite loss: Change at Day 268 | 0.00 (0.000)
  Appetite loss: Change at Day 296: number analyzed (Participants) | 2
  Appetite loss: Change at Day 296 | 16.67 (23.570)
  Appetite loss: Change at Day 324: number analyzed (Participants) | 1
  Appetite loss: Change at Day 324 | -33.33 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Constipation: Change at Day 7 | 0.00 (17.817)
  Constipation: Change at Day 28 | -4.17 (11.785)
  Constipation: Change at Day 56 | 0.00 (17.817)
  Constipation: Change at Day 78 | -4.17 (11.785)
  Constipation: Change at Day 100 | 0.00 (0.000)
  Constipation: Change at Day 128 | -4.17 (11.785)
  Constipation: Change at Day 156 | -4.17 (11.785)
  Constipation: Change at Day 184 | -4.17 (11.785)
  Constipation: Change at Day 212: number analyzed (Participants) | 6
  Constipation: Change at Day 212 | 0.00 (0.000)
  Constipation: Change at Day 240: number analyzed (Participants) | 3
  Constipation: Change at Day 240 | 0.00 (0.000)
  Constipation: Change at Day 268: number analyzed (Participants) | 2
  Constipation: Change at Day 268 | 16.67 (23.570)
  Constipation: Change at Day 296: number analyzed (Participants) | 2
  Constipation: Change at Day 296 | 50.00 (70.711)
  Constipation: Change at Day 324: number analyzed (Participants) | 1
  Constipation: Change at Day 324 | 0.00 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Diarrhea: Change at Day 7 | 8.33 (23.570)
  Diarrhea: Change at Day 28 | 0.00 (25.198)
  Diarrhea: Change at Day 56 | -12.50 (24.801)
  Diarrhea: Change at Day 78 | -12.50 (24.801)
  Diarrhea: Change at Day 100 | 0.00 (35.635)
  Diarrhea: Change at Day 128 | -8.33 (23.570)
  Diarrhea: Change at Day 156 | -8.33 (23.570)
  Diarrhea: Change at Day 184 | -8.33 (15.430)
  Diarrhea: Change at Day 212: number analyzed (Participants) | 6
  Diarrhea: Change at Day 212 | 0.00 (21.082)
  Diarrhea: Change at Day 240: number analyzed (Participants) | 3
  Diarrhea: Change at Day 240 | 11.11 (19.245)
  Diarrhea: Change at Day 268: number analyzed (Participants) | 2
  Diarrhea: Change at Day 268 | 33.33 (0.000)
  Diarrhea: Change at Day 296: number analyzed (Participants) | 2
  Diarrhea: Change at Day 296 | -16.67 (23.570)
  Diarrhea: Change at Day 324: number analyzed (Participants) | 1
  Diarrhea: Change at Day 324 | 33.33 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Financial difficulties: Change at Day 7 | -4.17 (21.362)
  Financial difficulties: Change at Day 28 | -4.17 (11.785)
  Financial difficulties: Change at Day 56 | -12.50 (17.252)
  Financial difficulties: Change at Day 78 | -8.33 (23.570)
  Financial difficulties: Change at Day 100 | -12.50 (17.252)
  Financial difficulties: Change at Day 128 | 0.00 (30.861)
  Financial difficulties: Change at Day 156 | -12.50 (17.252)
  Financial difficulties: Change at Day 184 | -12.50 (17.252)
  Financial difficulties: Change at Day 212 | -11.11 (27.217)
  Financial difficulties: Change at Day 240 | 0.00 (33.333)
  Financial difficulties: Change at Day 268 | -16.67 (23.570)
  Financial difficulties: Change at Day 296 | -16.67 (23.570)
  Financial difficulties: Change at Day 324 | -33.33 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.

31. Secondary Outcome: Phase 2: Change From Baseline in Patient Global Impression of Severity (PGIS) Score at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352, 380
Description: PGIS was a single item to assess severity of pain on a 5-point verbal rating scale ranged from 1 (no pain) to 5 (very severe pain), where 1: none; 2: mild; 3: moderate; 4: severe; 5: very severe. A higher score indicated a more severe pain.
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352, 380
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 54 | 8
Score on a scale
  Change at Day 7 | -0.3 (0.96) | 0.3 (0.71)
  Change at Day 28: number analyzed (Participants) | 52 | 8
  Change at Day 28 | -0.3 (0.94) | -0.1 (0.64)
  Change at Day 56: number analyzed (Participants) | 52 | 8
  Change at Day 56 | -0.3 (0.79) | 0.3 (0.46)
  Change at Day 78: number analyzed (Participants) | 46 | 8
  Change at Day 78 | -0.3 (0.87) | 0.0 (0.53)
  Change at Day 100: number analyzed (Participants) | 49 | 8
  Change at Day 100 | -0.3 (0.93) | 0.0 (0.53)
  Change at Day 128: number analyzed (Participants) | 40 | 8
  Change at Day 128 | -0.3 (1.06) | 0.0 (0.53)
  Change at Day 156: number analyzed (Participants) | 36 | 8
  Change at Day 156 | -0.4 (0.90) | 0.0 (0.93)
  Change at Day 184: number analyzed (Participants) | 39 | 8
  Change at Day 184 | -0.3 (1.06) | 0.3 (0.46)
  Change at Day 212: number analyzed (Participants) | 33 | 6
  Change at Day 212 | -0.2 (0.97) | 0.0 (0.63)
  Change at Day 240: number analyzed (Participants) | 31 | 3
  Change at Day 240 | -0.3 (0.86) | 0.0 (0.00)
  Change at Day 268: number analyzed (Participants) | 34 | 1
  Change at Day 268 | -0.5 (0.93) | 0.0 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was evaluated.
  Change at Day 296: number analyzed (Participants) | 33 | 2
  Change at Day 296 | -0.2 (1.20) | 0.0 (0.00)
  Change at Day 324: number analyzed (Participants) | 13 | 1
  Change at Day 324 | -0.6 (1.12) | 0.0 (NA) — Here, 'NA' signifies that SD could not be calculated as only 1 participant was analyzed.
  Change at Day 352: number analyzed (Participants) | 7 | 0
  Change at Day 352 | -0.9 (1.21) |
  Change at Day 380: number analyzed (Participants) | 2 | 0
  Change at Day 380 | -0.5 (0.71) |

32. Secondary Outcome: Phase 2: Patient Global Impression of Change (PGIC) Score at Days 28, 56, 78, 100
Description: PGIC was a single item to assess the participant's perception in change of their overall health status using a 7-point verbal rating scale ranging from 1(a lot better now) to 7 (a lot verse now), where 1: a lot better now; 2: moderately better now; 3: a little better now; 4: neither better nor worse; 5: a little worse now; 6: moderately worse now; 7: a lot worse now. Higher score indicated worse health status.
Time Frame: Days 28, 56, 78, 100
Population: mITT analysis set included all participants who received a JNJ-68284528 infusion at the targeted RP2D dose level. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 (US Population) | Phase 2 (Japan Population)
Number analyzed (Participants) | 54 | 8
Score on a scale
  Change at Day 28: number analyzed (Participants) | 52 | 8
  Change at Day 28 | 2.7 (1.63) | 2.8 (0.89)
  Change at Day 56 | 2.5 (1.66) | 2.9 (1.25)
  Change at Day 78: number analyzed (Participants) | 49 | 8
  Change at Day 78 | 2.2 (1.51) | 2.5 (0.93)
  Change at Day 100: number analyzed (Participants) | 54 | 7
  Change at Day 100 | 2.0 (1.43) | 2.4 (0.79)

33. Secondary Outcome: Phase 2 (US Population): Change From Baseline in EORTC QLQ-MY20 at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Description: EORTC QLQ-MY20 scale comprised of 20 questions that addressed four myeloma-specific HRQoL domains: disease symptoms (includes bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity), side effects of treatment (includes drowsiness, thirst, feeling ill, dry mouth, hair loss, upset by hair loss, tingling hands or feet, restlessness/agitation, acid indigestion/heartburn, and burning or sore eyes), future perspective (includes worry about death and health in the future, and thinking about illness) and body image. The scale was administered to assess 4 single items: feel restless or agitated, thinking about your illness, worried about dying, worried about health in the future. Scores were averaged and scales were transformed on a 0 to 100 scale. A high score for side effects of treatment represented a high level of symptomatology or problems, whereas a high score for future perspective represented better outcomes.
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296, 324, 352 and 380
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 54
Score on a scale
  Restless or agitated: Change at Day 7 | 5.7 [0.6 to 10.8]
  Restless or agitated: Change at Day 28: number analyzed (Participants) | 53
  Restless or agitated: Change at Day 28 | -5.5 [-10.7 to -0.3]
  Restless or agitated: Change at Day 56: number analyzed (Participants) | 52
  Restless or agitated: Change at Day 56 | 1.6 [-3.6 to 6.7]
  Restless or agitated: Change at Day 78: number analyzed (Participants) | 46
  Restless or agitated: Change at Day 78 | -2.7 [-8.1 to 2.8]
  Restless or agitated: Change at Day 100: number analyzed (Participants) | 49
  Restless or agitated: Change at Day 100 | -3.3 [-8.6 to 2]
  Restless or agitated: Change at Day 128: number analyzed (Participants) | 40
  Restless or agitated: Change at Day 128 | -3.9 [-9.6 to 1.9]
  Restless or agitated: Change at Day 156: number analyzed (Participants) | 36
  Restless or agitated: Change at Day 156 | 0.9 [-5 to 6.9]
  Restless or agitated: Change at Day 184: number analyzed (Participants) | 40
  Restless or agitated: Change at Day 184 | -3.6 [-9.4 to 2.1]
  Restless or agitated: Change at Day 212: number analyzed (Participants) | 33
  Restless or agitated: Change at Day 212 | -3.9 [-10.1 to 2.3]
  Restless or agitated: Change at Day 240: number analyzed (Participants) | 32
  Restless or agitated: Change at Day 240 | -12.7 [-19 to -6.5]
  Restless or agitated: Change at Day 268: number analyzed (Participants) | 35
  Restless or agitated: Change at Day 268 | -1.7 [-7.8 to 4.3]
  Restless or agitated: Change at Day 296: number analyzed (Participants) | 32
  Restless or agitated: Change at Day 296 | -7.8 [-14 to -1.5]
  Restless or agitated: Change at Day 324: number analyzed (Participants) | 14
  Restless or agitated: Change at Day 324 | -11.5 [-20.4 to -2.5]
  Restless or agitated: Change at Day 352: number analyzed (Participants) | 7
  Restless or agitated: Change at Day 352 | 1.1 [-11.1 to 13.4]
  Restless or agitated: Change at Day 380: number analyzed (Participants) | 2
  Restless or agitated: Change at Day 380 | -23.2 [-45.8 to -0.6]
  Thinking about illness: Change at Day 7 | 7.8 [1.7 to 14]
  Thinking about illness: Change at Day 28: number analyzed (Participants) | 53
  Thinking about illness: Change at Day 28 | 15 [8.8 to 21.2]
  Thinking about illness: Change at Day 56: number analyzed (Participants) | 52
  Thinking about illness: Change at Day 56 | 17.1 [10.8 to 23.3]
  Thinking about illness: Change at Day 78: number analyzed (Participants) | 46
  Thinking about illness: Change at Day 78 | 23.1 [16.7 to 29.6]
  Thinking about illness: Change at Day 100: number analyzed (Participants) | 49
  Thinking about illness: Change at Day 100 | 25.7 [19.4 to 32]
  Thinking about illness: Change at Day 128: number analyzed (Participants) | 40
  Thinking about illness: Change at Day 128 | 27.6 [20.8 to 34.3]
  Thinking about illness: Change at Day 156: number analyzed (Participants) | 35
  Thinking about illness: Change at Day 156 | 29.9 [22.8 to 36.9]
  Thinking about illness: Change at Day 184: number analyzed (Participants) | 40
  Thinking about illness: Change at Day 184 | 27.9 [21.2 to 34.7]
  Thinking about illness: Change at Day 212: number analyzed (Participants) | 33
  Thinking about illness: Change at Day 212 | 34.7 [27.5 to 41.8]
  Thinking about illness: Change at Day 240: number analyzed (Participants) | 32
  Thinking about illness: Change at Day 240 | 32.1 [24.8 to 39.3]
  Thinking about illness: Change at Day 268: number analyzed (Participants) | 35
  Thinking about illness: Change at Day 268 | 34.9 [27.8 to 41.9]
  Thinking about illness: Change at Day 296: number analyzed (Participants) | 32
  Thinking about illness: Change at Day 296 | 32.6 [25.3 to 39.8]
  Thinking about illness: Change at Day 324: number analyzed (Participants) | 14
  Thinking about illness: Change at Day 324 | 35.1 [25.3 to 45]
  Thinking about illness: Change at Day 352: number analyzed (Participants) | 7
  Thinking about illness: Change at Day 352 | 33.5 [20.3 to 46.8]
  Thinking about illness: Change at Day 380: number analyzed (Participants) | 2
  Thinking about illness: Change at Day 380 | 34.3 [10.2 to 58.4]
  Worried about dying: Change at Day 7 | 13.2 [8.5 to 17.8]
  Worried about dying: Change at Day 28: number analyzed (Participants) | 53
  Worried about dying: Change at Day 28 | 18.2 [13.6 to 22.9]
  Worried about dying: Change at Day 56: number analyzed (Participants) | 52
  Worried about dying: Change at Day 56 | 16.8 [12.1 to 21.5]
  Worried about dying: Change at Day 78: number analyzed (Participants) | 46
  Worried about dying: Change at Day 78 | 18.3 [13.4 to 23.1]
  Worried about dying: Change at Day 100: number analyzed (Participants) | 49
  Worried about dying: Change at Day 100 | 18.9 [14.1 to 23.7]
  Worried about dying: Change at Day 128: number analyzed (Participants) | 40
  Worried about dying: Change at Day 128 | 16.8 [11.7 to 21.9]
  Worried about dying: Change at Day 156: number analyzed (Participants) | 36
  Worried about dying: Change at Day 156 | 14.9 [9.6 to 20.2]
  Worried about dying: Change at Day 184: number analyzed (Participants) | 40
  Worried about dying: Change at Day 184 | 15.8 [10.7 to 21]
  Worried about dying: Change at Day 212: number analyzed (Participants) | 33
  Worried about dying: Change at Day 212 | 13.3 [7.9 to 18.8]
  Worried about dying: Change at Day 240: number analyzed (Participants) | 32
  Worried about dying: Change at Day 240 | 14.7 [9.1 to 20.2]
  Worried about dying: Change at Day 268: number analyzed (Participants) | 35
  Worried about dying: Change at Day 268 | 10 [4.7 to 15.4]
  Worried about dying: Change at Day 296: number analyzed (Participants) | 32
  Worried about dying: Change at Day 296 | 16.3 [10.8 to 21.8]
  Worried about dying: Change at Day 324: number analyzed (Participants) | 14
  Worried about dying: Change at Day 324 | 17.6 [9.9 to 25.3]
  Worried about dying: Change at Day 352: number analyzed (Participants) | 7
  Worried about dying: Change at Day 352 | 14.9 [4.5 to 25.3]
  Worried about dying: Change at Day 380: number analyzed (Participants) | 2
  Worried about dying: Change at Day 380 | 27.1 [8 to 46.1]
  Worried about health in future: Change at Day 7 | 8.2 [2.2 to 14.2]
  Worried about health in future: Change at Day 28: number analyzed (Participants) | 53
  Worried about health in future: Change at Day 28 | 18.2 [12.2 to 24.2]
  Worried about health in future: Change at Day 56: number analyzed (Participants) | 52
  Worried about health in future: Change at Day 56 | 15.5 [9.4 to 21.5]
  Worried about health in future: Change at Day 78: number analyzed (Participants) | 46
  Worried about health in future: Change at Day 78 | 19.7 [13.4 to 26]
  Worried about health in future: Change at Day 100: number analyzed (Participants) | 49
  Worried about health in future: Change at Day 100 | 14.3 [8.1 to 20.4]
  Worried about health in future: Change at Day 128: number analyzed (Participants) | 40
  Worried about health in future: Change at Day 128 | 20.4 [13.8 to 26.9]
  Worried about health in future: Change at Day 156: number analyzed (Participants) | 35
  Worried about health in future: Change at Day 156 | 18.9 [12 to 25.7]
  Worried about health in future: Change at Day 184: number analyzed (Participants) | 39
  Worried about health in future: Change at Day 184 | 19 [12.3 to 25.6]
  Worried about health in future: Change at Day 212: number analyzed (Participants) | 33
  Worried about health in future: Change at Day 212 | 19.9 [12.9 to 26.9]
  Worried about health in future: Change at Day 240: number analyzed (Participants) | 32
  Worried about health in future: Change at Day 240 | 19.7 [12.6 to 26.8]
  Worried about health in future: Change at Day 268: number analyzed (Participants) | 35
  Worried about health in future: Change at Day 268 | 17.1 [10.2 to 23.9]
  Worried about health in future: Change at Day 296: number analyzed (Participants) | 32
  Worried about health in future: Change at Day 296 | 24.2 [17.2 to 31.3]
  Worried about health in future: Change at Day 324: number analyzed (Participants) | 14
  Worried about health in future: Change at Day 324 | 20.2 [10.5 to 29.8]
  Worried about health in future: Change at Day 352: number analyzed (Participants) | 7
  Worried about health in future: Change at Day 352 | 25.1 [12.1 to 38]
  Worried about health in future: Change at Day 380: number analyzed (Participants) | 2
  Worried about health in future: Change at Day 380 | 7.7 [-15.8 to 31.2]

34. Secondary Outcome: Phase 2 (Japan Population): Change From Baseline in EORTC QLQ-MY20 at Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Description: as for outcome 33
Time Frame: Baseline, Days 7, 28, 56, 78, 100, 128, 156, 184, 212, 240, 268, 296 and 324
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 (US Population)
Number analyzed (Participants) | 8
Score on a scale
  Restless or agitated: Change at Day 7 | 12.50 (17.252)
  Restless or agitated: Change at Day 28 | 8.33 (15.430)
  Restless or agitated: Change at Day 56 | 0.00 (25.198)
  Restless or agitated: Change at Day 78 | 0.00 (17.817)
  Restless or agitated: Change at Day 100 | 0.00 (17.817)
  Restless or agitated: Change at Day 128 | 0.00 (25.198)
  Restless or agitated: Change at Day 156 | -8.33 (15.430)
  Restless or agitated: Change at Day 184 | -4.17 (21.362)
  Restless or agitated: Change at Day 212: number analyzed (Participants) | 6
  Restless or agitated: Change at Day 212 | -5.56 (13.608)
  Restless or agitated: Change at Day 240: number analyzed (Participants) | 3
  Restless or agitated: Change at Day 240 | -11.11 (19.245)
  Restless or agitated: Change at Day 268: number analyzed (Participants) | 2
  Restless or agitated: Change at Day 268 | -16.67 (23.570)
  Restless or agitated: Change at Day 296: number analyzed (Participants) | 2
  Restless or agitated: Change at Day 296 | 0.00 (0.000)
  Restless or agitated: Change at Day 324: number analyzed (Participants) | 1
  Restless or agitated: Change at Day 324 | -33.33 (NA) — SD could not be calculated as only 1 participant was analyzed.
  Thinking about illness: Change at Day 7 | 4.17 (33.034)
  Thinking about illness: Change at Day 28 | -4.17 (11.785)
  Thinking about illness: Change at Day 56 | 8.33 (15.430)
  Thinking about illness: Change at Day 78 | 4.17 (11.785)
  Thinking about illness: Change at Day 100 | 8.33 (15.430)
  Thinking about illness: Change at Day 128 | 8.33 (15.430)
  Thinking about illness: Change at Day 156 | 12.50 (24.801)
  Thinking about illness: Change at Day 184 | 12.50 (17.252)
  Thinking about illness: Change at Day 212: number analyzed (Participants) | 6
  Thinking about illness: Change at Day 212 | 22.22 (27.217)
  Thinking about illness: Change at Day 240: number analyzed (Participants) | 3
  Thinking about illness: Change at Day 240 | 0.00 (0.000)
  Thinking about illness: Change at Day 268: number analyzed (Participants) | 2
  Thinking about illness: Change at Day 268 | 0.00 (0.000)
  Thinking about illness: Change at Day 296: number analyzed (Participants) | 2
  Thinking about illness: Change at Day 296 | 0.00 (0.000)
  Thinking about illness: Change at Day 324: number analyzed (Participants) | 1
  Thinking about illness: Change at Day 324 | 0.00
  Worried about dying: Change at Day 7 | 16.67 (17.817)
  Worried about dying: Change at Day 28 | 8.33 (15.430)
  Worried about dying: Change at Day 56 | 16.67 (25.198)
  Worried about dying: Change at Day 78 | 25.00 (23.570)
  Worried about dying: Change at Day 100 | 25.00 (23.570)
  Worried about dying: Change at Day 128 | 25.00 (23.570)
  Worried about dying: Change at Day 156 | 20.83 (24.801)
  Worried about dying: Change at Day 184 | 29.17 (21.362)
  Worried about dying: Change at Day 212: number analyzed (Participants) | 6
  Worried about dying: Change at Day 212 | 27.78 (25.092)
  Worried about dying: Change at Day 240: number analyzed (Participants) | 3
  Worried about dying: Change at Day 240 | 11.11 (19.245)
  Worried about dying: Change at Day 268: number analyzed (Participants) | 2
  Worried about dying: Change at Day 268 | 16.67 (23.570)
  Worried about dying: Change at Day 296: number analyzed (Participants) | 2
  Worried about dying: Change at Day 296 | 16.67 (23.570)
  Worried about dying: Change at Day 324: number analyzed (Participants) | 1
  Worried about dying: Change at Day 324 | 0.00
  Worried about health in future: Change at Day 7 | 0.00 (17.817)
  Worried about health in future: Change at Day 28 | -4.17 (11.785)
  Worried about health in future: Change at Day 56 | 4.17 (21.362)
  Worried about health in future: Change at Day 78 | 4.17 (11.785)
  Worried about health in future: Change at Day 100 | 0.00 (0.000)
  Worried about health in future: Change at Day 128 | 0.00 (0.000)
  Worried about health in future: Change at Day 156 | 4.17 (11.785)
  Worried about health in future: Change at Day 184 | 8.33 (15.430)
  Worried about health in future: Change at Day 212: number analyzed (Participants) | 6
  Worried about health in future: Change at Day 212 | 5.56 (13.608)
  Worried about health in future: Change at Day 240: number analyzed (Participants) | 3
  Worried about health in future: Change at Day 240 | 22.22 (19.245)
  Worried about health in future: Change at Day 268: number analyzed (Participants) | 2
  Worried about health in future: Change at Day 268 | 0.00 (0.000)
  Worried about health in future: Change at Day 296: number analyzed (Participants) | 2
  Worried about health in future: Change at Day 296 | 0.00 (0.000)
  Worried about health in future: Change at Day 324: number analyzed (Participants) | 1
  Worried about health in future: Change at Day 324 | 0.00

ADVERSE EVENTS:
Time Frame: Day 1 up to 45.2 months
Description: All treated analysis set included all participants who received JNJ-68284528 infusion.
Arm/Group | Phase 1b (US Population) | Phase 2 (US Population) | Phase 2 (Japan Population)
All-Cause Mortality (participants affected / at risk) | 10/29 | 25/68 | 3/9
Serious Adverse Events (participants affected / at risk) | 11/29 | 42/68 | 1/9
Other Adverse Events (participants affected / at risk) | 29/29 | 68/68 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (US Population) (N=29) | Phase 2 (US Population) (N=68) | Phase 2 (Japan Population) (N=9)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Gait Disturbance (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 5 | 15 | 1
Atypical Pneumonia (Infections and infestations) | 1 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus Viraemia (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Cryptosporidial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lung Abscess (Infections and infestations) | 0 | 1 | 0
Perirectal Abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4 | 0
Rhinovirus Infection (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 4 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 0 | 0
Cranial Nerve Paralysis (Nervous system disorders) | 0 | 1 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0 | 0
Immune Effector Cell-Associated Neurotoxicity Syndrome (Nervous system disorders) | 1 | 4 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 2 | 0
Noninfective Encephalitis (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 3 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 3 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (US Population) (N=29) | Phase 2 (US Population) (N=68) | Phase 2 (Japan Population) (N=9)
Anaemia (Blood and lymphatic system disorders) | 22 | 57 | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 6 | 3
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 11 | 2
Leukopenia (Blood and lymphatic system disorders) | 20 | 40 | 4
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 16 | 35 | 0
Neutropenia (Blood and lymphatic system disorders) | 29 | 64 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 51 | 7
Sinus Bradycardia (Cardiac disorders) | 0 | 4 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 12 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 6 | 0
Constipation (Gastrointestinal disorders) | 7 | 14 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 19 | 2
Nausea (Gastrointestinal disorders) | 6 | 21 | 3
Vomiting (Gastrointestinal disorders) | 5 | 14 | 3
Asthenia (General disorders) | 3 | 2 | 0
Chills (General disorders) | 3 | 17 | 0
Fatigue (General disorders) | 6 | 30 | 1
Malaise (General disorders) | 2 | 1 | 1
Oedema Peripheral (General disorders) | 3 | 14 | 0
Pain (General disorders) | 2 | 2 | 0
Pyrexia (General disorders) | 2 | 17 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 26 | 59 | 7
Hypogammaglobulinaemia (Immune system disorders) | 1 | 11 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 4 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0
Rhinovirus Infection (Infections and infestations) | 2 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 6 | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 4 | 0
Alanine Aminotransferase Increased (Investigations) | 9 | 15 | 2
Aspartate Aminotransferase Increased (Investigations) | 10 | 18 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 10 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 12 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 11 | 1
International Normalised Ratio Increased (Investigations) | 1 | 8 | 0
Serum Ferritin Increased (Investigations) | 2 | 5 | 0
Weight Decreased (Investigations) | 3 | 2 | 0
Weight Increased (Investigations) | 2 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 25 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 8 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 21 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 29 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 17 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 12 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 20 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 24 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 11 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 9 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 10 | 0
Anosmia (Nervous system disorders) | 0 | 5 | 0
Dizziness (Nervous system disorders) | 4 | 14 | 0
Dysgeusia (Nervous system disorders) | 1 | 4 | 0
Headache (Nervous system disorders) | 5 | 14 | 3
Immune Effector Cell-Associated Neurotoxicity Syndrome (Nervous system disorders) | 2 | 11 | 0
Memory Impairment (Nervous system disorders) | 2 | 2 | 0
Micrographia (Nervous system disorders) | 0 | 4 | 0
Parosmia (Nervous system disorders) | 2 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 2 | 11 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 26 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 4 | 0
Embolism (Vascular disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 7 | 0
Hypertension (Vascular disorders) | 3 | 15 | 1
Hypotension (Vascular disorders) | 2 | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03548207/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03548207/SAP_001.pdf